

**Protocol Title:** Non-Invasive Brainstem Modulation for the Treatment of Non-Motor Symptoms in Parkinson's Disease: An Open Label Extension (OLE) Study: Statistical Analysis Plan (Brief Title: STEM-PD)

## STATISTICAL ANALYSIS PLAN

for OLE Study (ID: SNS-PD-003)

Protocol Version and Date: Version 6.0 (May 10, 2024)

Version 5.0 (February 15, 2023)

Version 4.0 (August 15, 2022)

Version 3.0 (December 14, 2021)

Version 2.0 (September 14, 2021)

Version 1.1 (May 17, 2021)

Version 1.0 (March 4, 2021)

# **Confidentiality Statement**

The information contained herein is confidential proprietary property of Scion NeuroStim, Inc. Any unauthorized use or disclosure of information expressed herein without the prior written authorization of Scion NeuroStim, Inc. is prohibited.

National Clinical Trial Identifiers: NCT04799418

List of authors and reviewers

Authors

Martin Slade, MPH, PhD, Lead Trial Statistician, Lecturer in Medicine, Lecturer in Public Health, Director of Research, Yale Occupational & Environmental Medicine

Kristen Ade, PhD, Vice President and Chief Scientific Officer, Scion NeuroStim, Inc.

Jennifer A. Elder, PhD, Chief Scientific Officer, PharPoint Research

## Reviewers

Robert Black, PhD, Chief Operating Officer and Chief Technology Officer, Scion NeuroStim, Inc.

Dawn Reilly-O'Dell, MPH, RAC, Lead Regulatory Consultant, Full Circle Regulatory Consulting, LLC

Ashley Weeks, MBiostat, Biostatistician II, PharPoint Research

# **Table of Contents**

| 1. | IN' | TRODUCTION | 5 |
|---|---|---|---|
| 2. | ST | UDY DESIGN | 5 |
| | 2.1. | STUDY OBJECTIVES | |
| | 2.2. | STUDY ENDPOINTS | 6 |
| <i>3</i> . | TR | EATMENT | 8 |
| 4. | SA. | MPLE SIZE DETERMINATION | 9 |
| <i>5</i> . | | TERIM ANALYSIS | |
| <b>6.</b> | IN | DEPENDENT DATA MONITORING | 9 |
| <i>7</i> . | ST | ATISTICAL METHODS | |
| | 7.1. | GENERAL METHODS | |
| | 7.2. | HANDLING DEPENDENT OBSERVATIONS | |
| | 7.3. | ANALYSIS POPULATIONS | 10 |
| | 7.4. | DEFINITIONS | 11 |
| | 7.5. | ANALYSIS OF STUDY CONDUCT | 12 |
| | 7.6. | DESCRIPTION OF THE DATASET USED FOR ANALYSIS | |
| | 7.7. | PARTICIPANT DISPOSITION | 13 |
| | 7.7. | 1. Demographics and Baseline Characteristics | 13 |
| | 7.7. | J | |
| | 7.7. | | |
| | <b>7.8.</b> | EFFICACY ANALYSIS | |
| | 7.8. | $\mathcal{I}$ | |
| | 7.8. | J 1 | |
| | 7.8. | $\boldsymbol{\mathcal{E}}$ | |
| | 7.8. | $\epsilon$ | |
| | | 2.2.1. Supportive Analysis: Clinical Significance | |
| | 7.8. | <i>y y</i> | |
| | 7.8. | 7 1 | |
| | 7.8.<br>7.8. | , | |
| | 7.8.<br>7.8. | | |
| | 7.8. | | |
| | 7.8. | | |
| | 7.9. | SAFETY ANALYSIS | |
| | 7.9 <b>.</b><br>7.9. | | |
| | 7.9.<br>7.9. | | |
| | 7.9 | | |

| 7 | 7.10. EXPLORATORY ANALYSES | | 18 |
|---|---|---|---|
| 7 | .11. AD | DITIONAL ANALYSES | 20 |
| | | Subgroup Analysis | 20 |
| 7 | .12. AD | DITIONAL SUPPORTING ANALYSES | 20 |
| | 7.12.1.1. | Supportive analysis to further explore clinical significance | 20 |
| | | Missing data | |
| 8. | REFER | ENCES | 22 |
| App | oendix 1: . | STEM-PD RCT SAP | 23 |

## 1. INTRODUCTION

This document describes the statistical analysis plan (SAP) for SNS-PD-003, the multicenter open label extension (OLE) study described in the protocol Non-Invasive Brainstem Modulation for the Treatment of Non-Motor Symptoms in Parkinson's Disease: A Randomized Controlled Trial (RCT) and an Open Label Extension (OLE) Study (Brief title: STEM-PD). This analysis plan is meant to supplement the study protocol and specifically refers to presentation of safety and efficacy analyses related to data collected through the first end of treatment (EOT1) period in the OLE on day 197 for the participants that received passive treatment during the RCT. Procedures related to SNS-PD-002, the preceding RCT study, are specified in a separate SAP (SAP v6.0 for RCT Study (ID: SNS-PD-002, NCT04797611), and the reader is referred to that document for all definitions of RCT specific measurements. Procedures related to exploratory analyses from SNS-PD-002 and SNS-PD-003, including data collected between days 197 and 365 in the OLE for the group that received passive treatment during the RCT and all OLE data for the group that received active treatment during the RCT, will be defined within appendices to this SAP. Any deviations from this analysis plan will be described in the clinical study report.

## 2. STUDY DESIGN

This is a single-arm open label extension to the multicenter, double-blind, placebo-controlled, pivotal clinical trial evaluating the safety and efficacy of twice daily time-varying caloric vestibular stimulation (tvCVS¹) treatments using a solid-state Device developed by Scion NeuroStim, Inc. (SNS), also known as ThermoNeuroModulation (TNM<sup>TM</sup>), for treating symptoms associated with Parkinson's disease (PD). The study will be conducted at 15 centers, at minimum, in the United States and the United Kingdom. The majority of centers will be in the United States. All of the participants randomized into the preceding double-blinded RCT who complete the required clinic visits will receive the opportunity to consent to participate in the OLE during which they will self-administer tvCVS treatments twice daily in the home setting over a period of 12 weeks (84 days), be followed during a 16 week (112 day) post-treatment follow-up period and then will self-administer tvCVS treatments twice daily in the home setting over an additional 8 week (56 day) period. Only participants that complete the RCT will be eligible to participate in the OLE. As such, there will be a maximum of 184 potential participants enrolled in the OLE, dependent on attrition in the RCT.

The proposed indication for use is for the treatment of symptoms of PD. For the RCT schedule of events, see the study protocol.

### 2.1. STUDY OBJECTIVES

**Primary Objective:** The primary objective is to further evaluate the effectiveness of the TNM<sup>TM</sup> Device treatments to reduce non-motor symptom burden in Parkinson's disease (PD) for the purposes of supporting reimbursement and clinical adoption.

<sup>&</sup>lt;sup>1</sup> tvCVS is the Scion NeuroStim - named method of applying caloric vestibular stimulation in a controlled, time-varying manner.

**Secondary Objectives:** This study will seek to further evaluate the effectiveness of TNM<sup>TM</sup> treatments to provide adjuvant therapeutic effectiveness beyond that observed with dopamine replacement therapies (DRTs) to (1) provide global improvements related to PD symptoms, (2) improve activities of daily living related to motor function, (3) provide clinically meaningful change (4) improve motor signs and symptoms and (5) improve quality of life (QoL) for participants with PD, for the purposes of supporting reimbursement and clinical adoption.

**Safety Objectives:** This study will seek to further establish the safety of TNM<sup>TM</sup> treatments by monitoring adverse event rates and further evaluating whether TNM<sup>TM</sup> is associated with a worsening of balance, functional mobility and gait in PD.

**Exploratory Objectives:** This study will seek to further establish the effectiveness of TNM<sup>TM</sup> therapy for treating specific non-motor symptoms (NMS) and in treating motor complications from dopamine replacement therapies. Outcomes will also further evaluate the clinical meaningfulness of symptomatic improvements and provide additional measures to support clinical adoption and establish the health economics of TNM<sup>TM</sup> as a therapy in PD. Patient-perceived effectiveness outcomes will also be evaluated through the Patient Global Impression of Improvement (PGI-I).

Other exploratory objectives that will not be covered in this SAP but rather will be covered in a separate statistical analysis plan include determination of whether increasing the length of the intervention increases the overall effectiveness or alters the safety of the intervention, determination of whether treatment effects of the intervention persist once the intervention is stopped, evaluation of the potential for disease-modifying properties of the intervention and determination of the effects of re-implementing the intervention after it had been stopped. Outcomes may also further explore the temporal kinetics of motor symptom response to treatment, further evaluate the potential of TNM<sup>TM</sup> treatments to improve gait and evaluate the relationship of treatment adherence to effectiveness and safety of the device, evaluate the of treatment to changes in body mass index, evaluate the temporal kinetics of treatment response for the MDS-NMS, MDS-UPDRS II, and the modified MDS-UPDRS part III, and evaluate the relationship of treatment to global improvement overall and non-motor function.

### 2.2. STUDY ENDPOINTS

## **Primary Endpoint**

• The change in the International Parkinson and Movement Disorder Society Nonmotor Rating Scale (MDS-NMS) total score<sup>1</sup>

## Secondary endpoints

- The change in the combined measure of The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale: Parts I, II and III
- The change in the International Parkinson and Movement Disorder Society Unified

Parkinson's Disease Rating Scale Part II: Motor Aspects of Experiences of Daily Living (MDS-UPDRS Part II) <sup>2</sup>

- The Overall Clinical Global Impressions Scale- Improvement (CGI-I)<sup>3</sup>
- The change in the International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III: Motor Exam (MDS-UPDRS Part III) <sup>2</sup>
- The change in the Parkinson's Disease Questionnaire 39 summary index score (PDQ-39SI)<sup>4</sup>

## Safety endpoints

- The change in the Mini Balance Evaluation Systems Test (mini-BESTest) total score<sup>5</sup>
- Adverse events (AEs) frequency

## **Exploratory endpoints**

## The change in:

- The Montreal Cognitive Assessment (MoCA)
- The Oral Symbol Digit Modality Test (oSDMT)
- The Modified Schwab and England Activities of Daily Living Scale (S&E)
- The Parkinson's Sleep Scale-2 (PDSS-2)
- The Epworth Sleepiness Scale (ESS)
- The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F)
- The Geriatric Depression Scale (GDS)
- The Parkinson's Anxiety Scale (PAS)
- The Patient Reported Outcomes in Parkinson's Disease (PRO-PD)
- The MDS-NMS Non-Motor Fluctuations (NMF) Total Score
- The Hoehn & Yahr score (H&Y)
- The Zarit Burden Interview (ZBI)
- Unified Parkinson's Disease Rating Scale Part I: Mentation, Behavior and Mood (UPDRS I)
- The Unified Parkinson's Disease Rating Scale Part IV: Complications of Therapy
- EncephaLog<sup>TM</sup> Finger Tapping Test (number of finger taps)
- EncephaLog<sup>TM</sup> Timed Up and Go Test (TUG)
  - 3-meter TUG (time to complete)
  - 10-meter TUG (stride length, cadence, rotation time, time to complete)
- The Patient Global Impression of Improvement (PGI-I)
- The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I: Non-Motor Aspects of Experiences of Daily Living (MDS-UPDRS Part I)
- Domains of the MDS-NMS
  - Depression
  - Anxiety
  - Apathy
  - Psychosis
  - Impulse control and related disorders
  - Cognition

- Orthostatic hypotension
- Urinary
- Sexual
- Gastrointestinal
- Sleep and wakefulness
- Pain
- Other

Treatment adherence and itemized answers from the following will be reported descriptively:

- a TNM<sup>TM</sup> Device usability survey
- The Unified Parkinson's Disease Rating Scale Part IV (UPDRS IV)

## 3. TREATMENT

All eligible study participants will self-administer active tvCVS treatments twice daily with the TNM<sup>TM</sup> Generation 4.0 Device during the first 112 days of the OLE (days 113-197 in the study protocol) and the last 56 days of the OLE (days 309-365 in the study protocol). There will be no treatments administered between the end of treatment 1 (EOT1) clinic visit on day 197 and the follow up 3 (FU3) clinic-visit on day 309.

## 4. SAMPLE SIZE DETERMINATION

Any of the 184 participants who randomize in the RCT and complete the RCT portion of the study will be eligible to participate in the OLE if they are able to consent to the OLE portion of the study. It is expected that approximately 166 participants (83 per RCT randomized group) will complete the RCT, and that there will be an additional 10% attrition. As a result, it is expected that 74 participants will make up the passive-active treatment group. This number is sufficient to detect a difference of 2.64 points in the MDS-UPDRS Part I total score for the null hypothesis that mean change scores for the passive-active treatment group at EOT1 in the OLE is equal to the mean change scores in the passive treatment group during the RCT and the alternative hypothesis that the mean change score of the passive-active treatment group at EOT1 in the OLE represents greater symptomatic improvement than that of the passive treatment group at the end of the RCT with a power of >98% given a mean difference of -2.64 and a standard deviation of 5.32 points and alpha of 0.05 for a paired t-test. Following the argument given in the RCT SAP (Appendix 1), this implies that the sample size should be sufficient to adequately power the highly correlated endpoint of MDS-NMS.

## 5. INTERIM ANALYSIS

No interim analysis is planned for the OLE.

## 6. INDEPENDENT DATA MONITORING

The TNM<sup>TM</sup> Device has been designated as a Non-Significant Risk Device for use in this study population. However, the Sponsor has chosen to implement an Independent Medical Monitor (IMM) for the preceding RCT and the OLE to provide independent safety monitoring and to confirm data integrity. The IMM is a physician with extensive experience in Parkinson's disease and clinical trials and has no perceived or real conflict of interest with the Sponsor or in the study outcomes. The IMM will review the research protocol and ongoing study activities with emphasis on data integrity, protocol adherence and study participant safety issues while making recommendations to the continuation, modification or conclusion of the trial. The IMM will review data at least four times per year during the RCT and OLE studies.

The Sponsor will also ensure critical safety and data points will be monitored per the STEM-PD Clinical Monitoring Plan (CMP) and the STEM-PD Data and Safety Management Plan (DSMP). A summary of key monitoring procedures is noted below:

Each site will be assigned a Clinical Research Associate (CRA) who will monitor the data to ensure the protection of rights and safety of human subjects, to verify the reported trial data are accurate, complete, and verifiable from source documents, and that the trial is conducted in compliance with the currently approved protocol/amendment(s), with Good Clinical Practice and with the applicable regulatory requirements. For all enrolled study participants, 100% source data review (SDR) and source data verification (SDV), where applicable, will occur of informed consent documents and process, inclusion and exclusion criteria, primary endpoints and key secondary endpoints (e.g., MDS-UPDRS Part III and CGI-I), all protocol deviations and safety reports, including adverse events and safety endpoints. Targeted source data verification will occur for all other endpoints per the Targeted Source Data Verification (TSDV) portion of the CMP. Review of study-wide trends and key risk indicator (KRI) metrics will be reviewed in a departmental meeting to occur at least once a month. If trends are identified, the Sponsor will review with the study-assigned medical monitor and implement a Correction and Preventative Action (CAPA) Plan. The study-specific Medical and Safety monitor, who has extensive experience with the device, will review and sign off on all AEs at least monthly, and all Unanticipated Adverse Device Effects (UADE) within 2 days of acknowledgment of the event. All UADEs will be reported to the ethics committees and all site Investigators per the protocol and regulatory requirements.

Previous studies with the Device have not reported any Serious Adverse Device Effects (SADEs) or UADEs. As none are anticipated for this study, if two or more serious and related adverse events (SADE or UADE) are reported, the study will pause while universality and unblinded review occurs by the Medical and Safety monitor. Additionally, the IMM is providing additional oversite for this study, and she/he will review these events for adjudication and agreement and will provide recommendations to the Sponsor.

## 7. STATISTICAL METHODS

## 7.1. GENERAL METHODS

Descriptive statistical methods will be used to summarize the data from this study, with formal hypothesis testing performed for the primary and key secondary efficacy endpoints. Unless stated

otherwise, the term "descriptive statistics" refers to number of participants, mean, median, standard deviation, minimum, and maximum for continuous data, and frequencies and percentages for categorical data. For categorical variables, the denominator of percentages will be the number of subjects in the treatment group, except for those collected by study visit and/or scheduled time point, in which case the denominator of percentages will be the number of subjects with a non-missing value at the visit and/or the scheduled time point.

All data collected during the study will be included in data listings. Unless otherwise noted, the data will be sorted first by RCT treatment group, subject number, and then by date within each subject number.

All statistical testing will be two-sided and will be performed using a significance (alpha) level of 0.05 unless otherwise specified. P-values will be presented to three decimal places. For exploratory endpoints, inferential analyses including 95% confidence intervals and p-values will be provided, and no statements about statistical significance will be made. The p-values will be provided as informational only.

The statistical analyses may be conducted with the SAS® software package version 9.4 or higher or with GraphPad Prism software version 9.3.1 or higher.

### 7.2. HANDLING DEPENDENT OBSERVATIONS

Due to the design of the OLE, a participant may have received treatment in a crossover nature. For those participants, special data handling methods are required. For the passive-active group, assessments will be assigned to the treatment received at the time of the given assessment. All observations captured up to the first treatment with active tvCVS will be assigned to the passive treatment. All observations at or after the first treatment with active tvCVS will be assigned to the active treatment.

### 7.3. ANALYSIS POPULATIONS

**Intent-to-treat Population (ITT):** All eligible participants who are allocated a device in the RCT and receive one treatment in the OLE will be included in the primary analysis of efficacy and safety.

Modified Intent to treat (mITT): All eligible participants who have completed at least one treatment with the study device allocated during the OLE and have completed at least one assessment during the OLE will be included in the mITT analysis. This will be considered a secondary analysis to supplement the findings of the primary analysis and will only be performed for endpoints for which regularly scheduled post-treatment data exists.

**Per-protocol Population (PP):** All eligible participants who (1) who demonstrate at least 70% treatment adherence with the Study Device during the first 12-week OLE treatment period, (2) have completed the regularly scheduled end of treatment period 1 visit (day 197), (3) have not had changes to medications used to treat motor and/or non-motor symptoms of PD between the baseline 1 (day 0) and OLE end of treatment period 1 visit (day 197) and (4) have not had changes

to medications that mimic motor and/or non-motor symptoms of PD between the baseline 1 (day 0) and OLE end of treatment period 1 visit (day 197) will be included in the PP analysis. This will be considered a secondary analysis to supplement the findings of the primary analysis and key secondary analyses.

#### 7.4. DEFINITIONS

**Study groups:** The group/cohort that originally received passive treatment during the RCT will be referred to as the passive-active group. The group/cohort that originally received active tvCVS treatment during the RCT will be referred to as the active-active group.

**Study day:** The study day will be calculated in reference to the date of the first baseline virtual visit during the RCT (Day 0). Although the informed consent for the OLE will be completed on day 113, plus or minus window days, because the RCT and OLE are part of the same protocol and the evaluation of effectiveness in the OLE depends on RCT data, all dates in this OLE SAP will be in reference to the first RCT visit (Day 0) as is specified in the protocol.

**Analysis day:** The analysis day will be calculated in reference to the date of the last assessment in RCT/first assessment in OLE (Day 113). Analysis day will be utilized for comparisons for passive-active participants.

**OLE Baseline value:** Values obtained at the End of Treatment (EOT) visit for the RCT will define the OLE baseline values. Values obtained at the most recent visit during the RCT will define the OLE baseline values in cases where data is missing for the EOT visit for the RCT.

**Adherence (%):** Adherence is defined as the total number of times subjects used the device in a given treatment period divided by twice the number of days the subject participated in that treatment period, multiplied by 100 to give a percentage.

**Duration of Follow-up:** The duration of follow-up will be defined as the number of days from the OLE Baseline until the End of Treatment period 2 (day 365) assessment or the last completed visit (phone call, virtual or in clinic).

#### **Adverse Event:**

Per protocol, an AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, users, or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device and the events related to the procedures involved. For purposes of analyses, any AE specified on the Adverse Events eCRF page is considered an AE.

### **Adverse Device Effect (ADE):**

Per protocol, an ADE is an AE related to the use of an investigational medical device. For purposes of analysis, any AE specified on the Adverse Events eCRF page that is possibly related, probably related, or related to the study device will be considered an ADE.

## **Serious Adverse Event (SAE):**

Per protocol, a SAE is an AE that has

- Led to death.
- Led to serious deterioration in the health of the participant, that either resulted in:
  - 1. A life-threatening illness or injury, or
  - 2. A permanent impairment of a body structure or a body function, or
  - 3. In-patient or prolonged hospitalization, or
  - 4. Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or body function.
- Led to fetal distress, fetal death or congenital abnormality or birth defect.

For analysis purposes, SAEs are AEs which are defined as serious on the Adverse Events eCRF.

## **Serious Adverse Device Effect (SADE):**

Per protocol, a SADE is an ADE that has resulted in any of the consequences characteristic of a serious adverse event. For analysis purposes, any AE on the Adverse Events eCRF page that is possibly related, probably related, or related to the study device and is noted as serious will be considered a SADE.

## **Unexpected Adverse Device Effect (UADE):**

Per protocol, a UADE is an SADE on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of participants. For analysis purposes, any event noted on the SADE/UADE Report eCRF page that is noted as a UADE will be considered a UADE.

SADEs and UADEs are AEs specified as such on the eCRF. More information on SAEs, ADEs, SADEs, and UADEs can be found in Protocol (Version 6.0: 02 Apr 2024) Section 8.2.

## 7.5. ANALYSIS OF STUDY CONDUCT

Descriptive statistics for the participants will be described for the ITT, mITT, and PP populations. Study treatment administration, duration of follow-up, discontinuation from study treatment and the reasons for discontinuation will be summarized. Coded protocol deviations and protocol violations will also be summarized as follows:

- Major/Important versus Minor versus No Impact, where:
  - Major/Important are protocol deviations that might significantly impact completeness, accuracy, and/or reliability of study data OR could significantly affect a participant's rights, safety or well-being
  - Minor are protocol deviations with minor impact on data quality or patient safety
  - No impact are protocol deviations that do not impact data quality or patient safety

## 7.6. DESCRIPTION OF THE DATASET USED FOR ANALYSIS

SAS-compatible and csv data sets will be exported directly from the iMediData RAVE Electronic Data Capture (EDC) platform. Exceptions may include data for the MDS-UPDRS Part III that has been re-scored by central blinded raters within the Machine Medicine Kelvin-PD platform, data related to Finger-tapping tests and Timed Up and Go tests captured with the Mon4t EncephaLog, treatment adherence data downloaded from the returned study Devices, a file that defines types of medications taken to address motor and nonmotor symptoms of PD including the levodopa equivalent daily dose for each participant, and a file that defines all the assignment of each consented participant into populations for analysis (e.g., ITT, mITT and PP) and reasons for exclusion and withdrawal where appropriate. Data for these exceptions will be provided as csv files created with Microsoft Excel.

### 7.7. PARTICIPANT DISPOSITION

Numbers of early withdrawals during the OLE will be reported descriptively overall and by treatment period, and categorized reasons provided for early withdrawal will be reported. Withdrawals due to similar adverse events will be grouped into categories.

### 7.7.1. Demographics and Baseline Characteristics

The following baseline characteristics at both the RCT baseline and the OLE baseline will be summarized for all participants for each analysis population (i.e., ITT, mITT and PP): age, sex, years since PD diagnosis, levodopa equivalent daily dose (LEDD) at start of treatment <sup>6</sup>, race and ethnicity.

Disease characteristics and motor phenotypes (i.e., tremor-dominant, postural instability gait difficulty or intermediate), postural instability and gait difficulty (PIGD) and Hoehn & Yahr scores will be reported and defined using methodology defined within the RCT (Appendix 1).

Comparability of baseline characteristics will be assessed. Here, these characteristics will be compared between the start of the RCT (during which time they would receive the passive

treatment) and the start of the OLE (during which time they will receive the active treatment). The characteristics will include disease characteristics, concomitant medications and outcome scores as these items may have changed over the course of the RCT. Descriptive statistics will be presented by corresponding timing of assessment (i.e., RCT Baseline or OLE Baseline). Differences in scores will be determined using a paired t-test or Wilcoxon Signed test for continuous variables and a McNemar's test for binary variables. Characteristics will be considered different in circumstances where p < 0.05. If baselines prove to be significantly different ( $\alpha = 0.05$ ), adjustments to corresponding efficacy analyses will be made by incorporating baseline level as a covariate.

### 7.7.2. Pre-study and Concomitant Medications

Within a group, the number and percentage of participants on concomitant therapies at RCT baseline and at the start of the OLE will be reported categorically using categories defined in section 7.6.3 of the SAP v6.0 for RCT Study (ID: SNS-PD-002).

Changes in medications to treat symptoms associated with PD during the RCT or the first 12-week treatment period of the OLE are protocol deviations. As such, changes in these medications would exclude participants from the PP analysis. Changes in medications in the mITT and the ITT populations will be summarized descriptively.

Certain concomitant medications (e.g., antihistamines or acetylcholinesterase inhibitors) may alter treatment efficacy by affecting neurotransmitter systems involved in the mechanisms of action for tvCVS. Subgroup analyses will be performed to compare treatment effects in study participants taking these concomitant medications during the trial.

### 7.7.3. Study Device Administration

Treatment adherence will be analyzed for the OLE. Treatment adherence data will be reported descriptively. Treatment adherence  $\geq 70\%$  during the first 12-week treatment period in the OLE will be required for inclusion in the PP analysis (see section 7.2).

### 7.8. EFFICACY ANALYSIS

<sup>7</sup>Analysis of continuous endpoints will be conducted utilizing the methodology as described in section 7.7 of the SAP v6.0 for RCT Study (Appendix 1). For comparisons within the passive-active arm, the visit variable will be based on the adjusted analysis visit for the active comparisons and the subject effect of the model will be nested within ARM to account for the crossover nature of these data. For efficacy endpoints that have a baseline defined, only participants who have baseline data collected for the endpoints will be included in efficacy analyses.

## 7.8.1. Primary Objectives:

The primary objective is to further evaluate the effectiveness of TNM<sup>TM</sup> Device treatments to reduce non-motor symptom burden in PD for the purposes of supporting reimbursement and clinical adoption.

### 7.8.2. Primary Endpoint and Comparison of Interest

The primary endpoint is the change in MDS-NMS total score at the end of treatment. The primary comparison is its change in MDS-NMS total score during the RCT treatment period (days 29-113) versus the change in MDS-NMS total score during the OLE treatment period 1 (days 113-197). This analysis of the primary comparison will only utilize the passive-active treatment group. The analysis will utilize data obtained during the RCT as well as data obtained from the OLE baseline and the twelve weeks of the OLE in which the participants will have been given the intervention.

## 7.8.2.1. Statistical Significance

The null hypothesis is that 12 weeks of active tvCVS treatments during the OLE will yield an equivalent change in the passive-active treatment group of NMS burden as that which occurred in response to passive treatment during the RCT. The alternative hypothesis is that the passive-active treatment group will demonstrate a greater reduction of NMS burden after 12 weeks of active tvCVS treatment during the OLE than occurred after 12 weeks of passive treatment during the RCT. Rejection of the null hypothesis will indicate that the intervention was successful. The threshold to determine statistical significance will be set at  $\alpha = 0.05$  based upon a 1-tailed test.

## 7.8.2.2. Clinical Significance

Clinical significance is defined by how a treatment affects the extent to which a subject is currently living independent of help from others OR that there is a real genuine, palpable, and noticeable effect on daily life or how a patient feels, functions, or survives. Importantly, as the scores from the MDS-NMS are derived from the product of the symptom frequency (how often the patient has experienced a given non-motor symptom since the last evaluation with higher scores indicating more frequent experience) and symptom severity (impact of that symptom on how the patient has felt and functioned with higher scores indicating greater distress or disturbance to patient or caregiver), reductions in MDS-NMS total scores are inherently clinically meaningful in that they indicate improvements in how the participant is feeling and functioning. Given the inherent clinical meaningfulness of the MDS-NMS total score, the primary endpoint will be considered clinically meaningful, and therefore, successful, if there are statistically significant reductions in MDS-NMS total scores after active tvCVS treatment during the OLE relative to the change in response to the 12 weeks of passive treatment during the RCT.

## 7.8.2.2.1. Supportive Analysis: Clinical Significance

Data collected during the RCT will be used to define a Minimally Important Clinical Difference (MCID) in the primary outcome measure (the MDS-NMS).

Supportive analyses will also be conducted on the data from the OLE to determine whether the difference in the change scores between the active treatment in the OLE and the passive treatment during the RCT exceeds the MCID defined for the MDS-NMS in the RCT. This test will be based on the MMRM model described in Section 7.7 of the RCT SAP (Appendix 1), comparing the least-squares mean change of the active treatment (as estimated by the model) to the point estimate of the MCID determined from the RCT.

## 7.8.3. Secondary Objectives:

This study will seek to further evaluate the effectiveness of TNM<sup>TM</sup> treatments to provide adjuvant therapeutic effectiveness beyond that observed with DRTs to (1) provide global improvements related to PD symptoms, (2) improve activities of daily living related to motor function, (3) provide clinically meaningful change (4) improve motor symptoms and (5) improve quality of life (QoL) for participants with PD, for the purposes of supporting reimbursement and clinical adoption.

### 7.8.4. Secondary Endpoints

Multiplicity of study endpoints will be adjusted for using a hierarchical strategy whereby endpoints in the study are only considered to be statistically significant if both of the following are true: 1) p < 0.05 <u>AND</u> 2) the preceding endpoint was found to be statistically significant at the significance level  $\alpha = 0.05$ . More specifically, the hierarchical order for evaluation of efficacy endpoints is the following:

- 1. MDS-NMS Total Score (primary endpoint);
- 2. Combined measure of MDS-UPDRS Parts I, II, and III (sum score)
- 3. MDS-UPDRS Part II (secondary endpoint);
- 4. Overall CGI-I (secondary endpoint);
- 5. MDS-UPDRS Part III (secondary endpoint);
- 6. PDQ-39SI (secondary endpoint).

Note that all secondary endpoints have an *a priori* direction, thus, one-tailed tests will be utilized for analyses.

Secondary endpoint analysis will be conducted using the passive-active treatment group for the primary comparison of interest.

Analyses of the secondary endpoints will be conducted in a manner consistent with the primary endpoint except where noted.

#### 7.8.4.1. Combined measure of MDS-UPDRS Parts I, II, and III (sum score)

This endpoint will evaluate the change in the combined measure of MDS-UPDRS Parts I, II and III. The combined measure of MDS-UPDRS Parts I, II, III will be calculated, inclusive of imputation, as described in SAP v6.0 for RCT Study (Appendix 1). For the passive-active group, the change from corresponding baseline to end of treatment

period will be evaluated using a MMRM model similar to the one described for the primary analysis. Treatment differences will be assessed based on the least-squares mean change scores between the passive and active treatments. Changes meeting or exceeding the previously established MCID for this measure (-6.7 points for clinical improvement)<sup>8</sup> will be considered clinically meaningful.

### 7.8.4.2. MDS-UPDRS Part II

This endpoint will evaluate the change in MDS-UPDRS Part II score to provide a measure of activities of daily living related to motor function. The total score for MDS-UPDRS Part II will be calculated as described in the SAP v6.0 for RCT Study (Appendix 1). For the passive-active group, the change from corresponding baseline to end of treatment period will be evaluated using a MMRM model similar to the one described for the primary analysis. Treatment differences will be assessed based on the least-squares mean change scores between the passive and active treatments. Changes will be considered to be clinically meaningful if the mean difference exceeds the previously established MCID (-3.05 for clinical improvement)<sup>9</sup>.

#### 7.8.4.3. Overall CGI-I

The CGI-I provides a clinician's determination of overall change as it relates to all aspects of Parkinson's disease. For ease of interpretation, the CGI-I score will be converted by the following formula: Converted CGI-I = 4 – CGI-I. Thus a 0 corresponds to no change, higher magnitude positive values correspond to greater improvements and higher magnitude negative scores correspond to increased worsening. For the passive-active group, treatment differences will be modeled utilizing the MMRM with no effect for visit as described previously. The effect of the device in the OLE will be considered clinically significant if converted CGI-I scores after active tvCVS during the OLE are statistically significantly greater to those after passive treatment in the RCT.

#### 7.8.4.4. MDS-UPDRS Part III

The change in MDS-UPDRS Part III total score provides a measure of impact on motor signs in PD. This endpoint will be constructed, inclusive of imputation, as described in SAP v6.0 for RCT Study (Appendix 1). For the passive-active group, primary comparisons will be constructed using the MMRM model as previously described. Changes will be considered to be clinically meaningful if the mean difference exceeds the previously established MCID (-3.25 for clinical improvement) for this scale<sup>10</sup>.

## 7.8.4.5. PDQ-39SI

The PDQ39-SI will be calculated as described in the SAP v6.0 for RCT Study (Appendix 1). For the passive-active group, primary comparisons will be constructed using the MMRM model as previously described. Changes will be considered to be clinically meaningful if the mean difference exceeds the previously established MCID (-4.72 for clinical improvement) for this scale<sup>11</sup>.

### 7.9. SAFETY ANALYSIS

### 7.9.1. Adverse Events (AEs)

Participants will be assessed for AEs every two weeks at minimum (either at study visits or during phone calls). For each group, the AEs will be summarized with frequency and percentage by preferred (PT) term, with all participants in that treatment group as the denominator. Classification will utilize MedDRA System Organ Class (SOC) based on MedDRA® Version 26.0 or other terminology/classification common to Parkinson's disease (e.g., falls, freezing of gait, etc.). AE incidence will be summarized by both severity and causal relationship to Device treatment (as determined by the blinded Principal Investigator or designated study personnel). AEs deemed to be of "possible" or "probable" relationship or "related" to the Device will also be considered as device related. AEs that occurred during the baseline period and post randomization will also be summarized. Additionally, the number of events and number of device-related events per person will be reported as a distribution.

The AE summary tables will provide an overall summary of AEs including the number and percentage of participants who experienced any AE, any SAE, any ADE, any SADE, any UADE, and any discontinuations in study participation due to an AE.

The objectives for the adverse event analysis in this study will be to confirm the safety/tolerability of tvCVS for the treatment of PD. For this, AE rates will be evaluated in the passive-active cohort. McNemar's test will be used to compare AE rates with tvCVS treatment during the first 12-week treatment period of the OLE as compared to AE rates during the passive treatment period in the RCT. Examination of the safety/tolerability of treatment periods longer than 12-weeks, will be evaluated as part of the procedures described within the appendices to this SAP.

### 7.9.2. Safety Endpoint

The change in the mini-BESTest will serve as an additional safety endpoint to confirm that TNM<sup>TM</sup> treatment does not negatively impact balance in PD. Mini-BESTest data collected in the OFF-state will not be included in any analysis. <sup>12</sup>For the passive-active cohort, two sided, 95% confidence intervals for the Mini-BESTest median change score will be constructed difference between the for the passive treatment (RCT) and the tvCVS treatment (OLE) treatment period. If upper bound of the 95% confidence interval is less than 4 <sup>13</sup> then the no clinically meaningful difference between the groups exists.

### 7.10. EXPLORATORY ANALYSES

These exploratory endpoints have been added to support clinical applicability of the primary and secondary endpoints. They have been selected to provide additional detail that will impact decisions made by prescribing physicians and reimbursement entities.

Changes from baseline in the following assessments will be evaluated:

- 1. The Montreal Cognitive Assessment (MoCA)
- 2. The oral Symbol Digit Modality Test (oSDMT)
- 3. The Modified Schwab & England Activities of Daily Living Scale (S&E)
- 4. The Parkinson's Disease Sleep Scale-2 (PDSS-2)
- 5. The Epworth Sleepiness Scale (ESS)
- 6. The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F)
- 7. The Geriatric Depression Scale (GDS)
- 8. The Parkinson's Anxiety Scale (PAS)
- 9. The Patient Reported Outcome Parkinson's Disease (PRO-PD). The PRO-PD collected at the study screen will be used as a practice-only and will not be included in the analysis as the scale's author has indicated that scores from the first completion of the assessment typically have high variability relative to the scores from subsequent administrations.
- 10. The MDS-NMS Non-Motor Fluctuations (NMF) Total Score
- 11. The Hoehn & Yahr score (H&Y)
- 12. Zarit Burden Interview (ZBI)
- 13. The Unified Parkinson's Disease Rating Scale Part I (UPDRS I)
- 14. The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I: Non-Motor Aspects of Experiences of Daily Living (MDS-UPDRS Part I)
- 15. EncephaLog<sup>TM</sup> Finger Tapping Test the RCT baseline for this outcome will be the mean of scores collected weekly between Day 0 and Day 28.
- 16. EncephaLog<sup>TM</sup> 3m Timed Up and Go Test (3m TUG) Test the RCT baseline for this outcome will be the mean of scores collected weekly between Day 0 and Day 28.
- 17. EncephaLog<sup>TM</sup> 10m Timed Up and Go Test (10m TUG) This endpoint will evaluate the change in several measures related to the conduct of the 10-meter TUG at the end of the treatment period (day 113) relative to the baseline (day 29) including stride length, cadence, rotation time and time to complete.

For the primary comparison of interest (i.e. passive-active group following 12 weeks of treatment), the least-squares mean differences with corresponding 95% confidence intervals and p values will be constructed using the MMRM model discussed previously. However, no regulatory claims will be made in relation to these outcomes. Therefore, no adjustments will be made to address multiplicity of endpoints.

Treatment adherence, the Patient Global Impression of Improvement (PGI-I) and itemized answers from both the TNM<sup>TM</sup> Useability Questionnaire and the UPDRS IV assessment tool for the passive-active group will be reported descriptively. To further explore the effects of treatment on individual NMS, effects of treatment on each of the individual MDS-NMS domains will be evaluated. These domains include the following: (1) Depression, (2) Anxiety, (3) Apathy, (4) Psychosis, (5) Impulse control and related disorders, (6) Cognition, (7) Orthostatic hypotension, (8) Urinary, (9) Sexual, (10) Gastrointestinal, (11) Sleep and wakefulness, (12) Pain, and (13) Other. Only participants that demonstrate burden in the specified domain will be evaluated. In practice, this means that if any participant shows no burden on a given MDS-NMS domain throughout the study, then they will be excluded from this exploratory analysis.

### 7.11. ADDITIONAL ANALYSES

## 7.11.1. Subgroup Analysis

An analysis of the primary endpoint and select secondary endpoints will be conducted by country to determine if there is a different treatment effect in the United Kingdom as compared to the United States. For this analysis, separate models will be constructed per subgroup.

Other primary endpoint and select secondary endpoint subgroups to be evaluated include: Sponsor name utilized in ICF (Sponsor name in ICF vs Sponsor not in ICF), Prohibited Concomitant Medication Use (Used vs Not Used), the subset of confounding protocol deviations as noted in section 7.10.3 of the RCT SAP (see Appendix 1), specifically, a change in medication that mimics symptoms of Parkinson's disease occurred, a change in medication used to treat motor and/or non-motor symptoms of Parkinson's disease occurred and/or data was collected at a visit performed out of window when the participant was not treating when protocol requires (Present, Not Present).

### 7.12. ADDITIONAL SUPPORTING ANALYSES

## 7.12.1.1. Supportive analysis to further explore clinical significance

Although the structure and methodology for data collection of the MDS-NMS allows for interpretation of the statistically significant changes to be interpreted as inherently clinically meaningful, the scale is relatively new and not well known. As such, to support future clinical adoption by referring physicians, a supplementary analysis is planned as part of the procedures specified in the Statistical Analysis Plan for SNS-PD-002 to establish the MCID for the MDS-NMS. The MCID value identified in the analysis for SNS-PD-002 will define the MCID for analysis in these supporting analyses.

To support the clinical significance of the primary endpoint, the responder rate (i.e., percentage that demonstrate change scores during the first treatment period of the OLE ≥ the MCID) in the passive-active treatment group will be reported. Additionally, a McNemar's test will be employed to determine if the responder rate is statistically significantly greater after 12 weeks of tvCVS treatment during the OLE than was the responder rate for this group after 12 weeks of passive treatment during the RCT. The required percentage of participants during the OLE tvCVS that demonstrate a change exceeding the MCID to be statistically significant will be a function of the percentage of participants in the passive-active treatment group that demonstrate a change exceeding the MCID after passive treatment during the RCT. This relationship is depicted in Figure 2. Because the power of this binomial comparison will be reduced under conditions where there is a high responder rate of passive treatment participants during the RCT, if 36% or more of the RCT passive treatment group exceeds the MCID (a condition that would require > 60% responder rate in the active group), the clinical significance for the primary outcome measure will be established by verifying that the

mean difference between responses to the passive treatment RCT and the tvCVS treatment in the OLE exceeds the change equivalent to the MCID.





**Percent of Placebo Group Exceeding MCID** 

Figure 1: Effect of Percent in Passive (i.e., aka placebo or inactive) Group Exceeding MCID.

## 7.13. Missing data

Item-level missing data will be handled as described in the SAP v6.0 for RCT Study (ID: SNS-PD-002).

#### 8. REFERENCES

- 1. Chaudhuri KR, Schrag, A., Weintraub, D., Rizos, A., Rodriguez-Basquez, C., Mamikonyan, E., Martinez-Martin, P. The Movement Disorder Society Nonmotor Rating Scale: Initial Validation Study. Movement Disorders 2020;35:17.
- 2. Goetz CG, Tilley BC, Shaftman SR, et al. Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results. Mov Disord 2008;23:2129-2170.
- 3. Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont) 2007;4:28-37.
- 4. Jenkinson C, Fitzpatrick R, Peto V, Greenhall R, Hyman N. The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score. Age Ageing 1997;26:353-357.
- 5. Bloem BR, Marinus J, Almeida Q, et al. Measurement instruments to assess posture, gait, and balance in Parkinson's disease: Critique and recommendations. Mov Disord 2016;31:1342-1355.
- 6. Jost ST, Kaldenbach MA, Antonini A, et al. Levodopa Dose Equivalency in Parkinson's Disease: Updated Systematic Review and Proposals. Mov Disord 2023;38:1236-1252.
- 7. Rubin DB, & Schenker, N. Interval estimation from multiply-imputed data: a case study using census agriculture industry codes. Journal of Official Statistics 1987;3:375.
- 8. Makkos A, Kovacs M, Aschermann Z, et al. Are the MDS-UPDRS-Based Composite Scores Clinically Applicable? Mov Disord 2018;33:835-839.
- 9. Horvath K, Aschermann Z, Kovacs M, et al. Minimal clinically important differences for the experiences of daily living parts of movement disorder society-sponsored unified Parkinson's disease rating scale. Mov Disord 2017;32:789-793.
- 10. Horvath K, Aschermann Z, Acs P, et al. Minimal clinically important difference on the Motor Examination part of MDS-UPDRS. Parkinsonism Relat Disord 2015;21:1421-1426.
- 11. Horvath K, Aschermann Z, Kovacs M, et al. Changes in Quality of Life in Parkinson's Disease: How Large Must They Be to Be Relevant? Neuroepidemiology 2017;48:1-8.
- 12. Godi M, Franchignoni F, Caligari M, Giordano A, Turcato AM, Nardone A. Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders. Phys Ther 2013;93:158-167.
- 13. Ganju J, Rom D. Non-inferiority versus superiority drug claims: the (not so) subtle distinction. Trials 2017;18:278.

9.0 APPENDICES

Appendix 1: STEM-PD RCT SAP

**Protocol Title:** Non-Invasive Brainstem Modulation for the Treatment of Non-Motor Symptoms in Parkinson's Disease: A Randomized Controlled Trial (RCT): Statistical Analysis Plan (Brief Title: STEM-PD)

## STATISTICAL ANALYSIS PLAN v6.0

for RCT Study (ID: SNS-PD-002)

### **Protocol Version and Date:**

Version 6.0 (May 10, 2024)

Version 5.0 (February 15, 2023)

Version 4.0 (August 15, 2022)

Version 3.0 (December 14, 2021)

Version 2.0 (September 14, 2021)

Version 1.1 (May 17, 2021)

Version 1.0 (March 4, 2021)

# **Confidentiality Statement**

The information contained herein is confidential proprietary property of Scion NeuroStim, Inc. Any unauthorized use or disclosure of information expressed herein without the prior written authorization of Scion NeuroStim, Inc. is prohibited.

List of authors and reviewers

Authors

Martin Slade, MPH, PhD, Lead Trial Statistician, Lecturer in Medicine, Lecturer in Public Health, Director of Research, Yale Occupational & Environmental Medicine

Kristen Ade, PhD, Vice President and Chief Scientific Officer, Scion NeuroStim, Inc.

Jennifer A. Elder, PhD, Chief Scientific Officer, PharPoint Research

### Reviewers

Dawn Reilly-O'Dell, MPH, RAC, Lead Regulatory Consultant, Full Circle Regulatory Consulting, LLC

Robert Black, PhD, Chief Operating Officer and Chief Technology Officer, Scion NeuroStim, Inc.

Kara Richardson, Vice President of Clinical Affairs, Scion NeuroStim, Inc.

Ashley Weeks, MBiostat, Biostatistician II, PharPoint Research

# **Table of Contents**

| <i>1</i> . | INT | RODUCTION | 5 |
|---|---|---|---|
| 2. | STU | UDY DESIGN | 5 |
| 2 | 2.1. | STUDY OBJECTIVES | |
| | 2.2. | STUDY ENDPOINTS | |
| <i>3</i> . | | NDOMIZATION AND BLINDING | |
| | | MPLE SIZE DETERMINATION | |
| <i>4</i> . | | | |
| <i>5</i> . | NO | N-COMPARATIVE INTERIM ANALYSIS | 9 |
| <b>6.</b> | IND | DEPENDENT DATA MONITORING | 12 |
| <i>7</i> . | <b>ST</b> A | TISTICAL METHODS | 12 |
| , | 7.1. | GENERAL METHODS | 13 |
| , | 7.2. | ANALYSIS POPULATIONS | |
| | 7.3. | DEFINITIONS | |
| | 7.4. | ANALYSIS OF STUDY CONDUCT | |
| | 7.5. | DESCRIPTION OF THE DATASET USED FOR ANALYSIS | |
| • | <b>7.6.</b><br>7.6.1 | ANALYSIS OF TREATMENT GROUP COMPARABILITY Demographics and Baseline Characteristics | |
| | 7.6.1 | | |
| | 7.6.2 | | |
| | 7.6.4 | • | |
| • | 7.7. | EFFICACY ANALYSIS | 18 |
| | 7.7.1 | . Primary Endpoint | 20 |
| | 7.7.1 | $\varepsilon$ | |
| | 7.7.1 | č | |
| | 7.7.1 | | |
| | 7.7.2 | • • | |
| | 7.7.2<br>7.7.2 | , | |
| | 7.7.2 | | |
| | 7.7.2 | | |
| , | 7 <b>.8.</b> | SAFETY ANALYSIS | 28 |
| | 7.8.1 | . Adverse Events (AEs) | 28 |
| | 7.8.2 | | |
| , | 7.9. | EXPLORATORY ANALYSES | 28 |
| , | 7.10. | ADDITIONAL SENSITIVITY ANALYSES | 30 |
| | 7.10 | 1 Item level Missing Data | 30 |

| 7.10 | 0.2. Missing data | 32 |
|-------|----------------------------------------|----|
| 7.10 | | |
| 7.10 | | 3 |
| 7.10 | | 32 |
| 7.10 | 0.6. Physical limitations | 32 |
| 7.10 | 0.7. Country and Other Subgroups | 32 |
| 7.10 | | |
| 7.11. | ADDITIONAL SUPPORTING ANALYSES | 33 |
| 8. RE | FERENCES | 34 |
| 9. AP | PPENDICES | |
| Appen | ndix 1: STEM-PD RCT Schedule of Events | 37 |
| STEM | | |

## 1. INTRODUCTION

This document describes the statistical analysis plan (SAP) for SNS-PD-002, the multicenter randomized controlled trial portion described in the protocol Non-Invasive Brainstem Modulation for the Treatment of Non-Motor Symptoms in Parkinson's Disease: A Randomized Controlled Trial (RCT) and an Open Label Extension (OLE) Study (Brief title: STEM-PD). This analysis plan is meant to supplement the study protocol and specifically refers to procedures related to the RCT. Additional exploratory procedures of RCT data as well as procedures related to SNS-PD-003, the subsequent OLE portion of the study, will be specified in a separate SAP or Addendum. Any deviations from this analysis plan will be described in the clinical study report.

## 2. STUDY DESIGN

This is a randomized (1:1), multicenter, double-blind, controlled, pivotal clinical trial evaluating the safety and efficacy of twice daily time-varying caloric vestibular stimulation (tvCVS<sup>1</sup>) treatments using a solid-state Device developed by Scion NeuroStim, Inc. (SNS), also known as ThermoNeuroModulation (TNMTM), for treating symptoms associated with Parkinson's disease (PD). The study will be conducted at 15 centers, at minimum, located in either the United States or the United Kingdom. The majority of centers will be in the United States. Up to 290 participants will screen for the randomized clinical trial (RCT) and will self-administer either tvCVS treatments or passive treatments twice daily in the home setting over a period of 12 weeks (84 days). Participants will continue to be enrolled into the RCT until at least 184 participants have randomized at which point competitive enrollment will be closed. The RCT will be immediately followed by an open label extension (OLE) study. The RCT and OLE have been separated into two distinct portions of the study with separate informed consent to enable the closeout and analysis of the RCT portion which will support regulatory submissions during the conduct of the OLE. However, anticipated participation in the OLE study will be a selection criterion for participating in the RCT, and thus, the two studies are defined within the context of a single protocol.

The proposed indication for use is for the treatment of symptoms of PD. For the RCT schedule of events, see <u>Appendix 1</u>.

### 2.1. STUDY OBJECTIVES

The null hypothesis for each of the primary and secondary outcomes states that the two treatment groups will show an equivalent change after 12 weeks of twice daily treatment with the TNM<sup>TM</sup> Device.

<sup>&</sup>lt;sup>1</sup> tvCVS is the Scion NeuroStim - named method of applying caloric vestibular stimulation in a controlled, time-varying manner.

**Primary Objectives:** The primary objective of the RCT will be to test the hypothesis that TNM<sup>TM</sup> treatments provide safe and effective therapy for the reduction of non-motor symptom burden in participants with PD.

**Secondary Objectives:** This study will seek to establish whether TNM<sup>TM</sup> treatments provide adjuvant therapeutic effectiveness beyond that observed with dopamine replacement therapies (DRTs) to (1) provide global improvements, (2) improve activities of daily living related to motor function, (3) provide clinically meaningful change, (4) improve motor signs and symptoms and (5) improve quality of life (QoL) for participants with PD.

**Safety Objectives:** This study will seek to establish the safety of TNM<sup>TM</sup> by monitoring adverse events and evaluating whether TNM<sup>TM</sup> is associated with a worsening of balance, functional mobility and gait in PD.

**Exploratory Objectives:** This study will seek to establish the effectiveness of TNM<sup>TM</sup> treatments for reducing specific non-motor symptoms (NMS) and in treating motor complications of dopamine replacement therapies. Outcomes will also evaluate the clinical meaningfulness of symptomatic improvements, explore the temporal kinetics of motor symptom response to treatment, evaluate the potential of TNM<sup>TM</sup> treatments to improve gait, and provide additional measures to support clinical adoption and establish the health economics of TNM<sup>TM</sup> as a therapy in PD.

#### 2.2. STUDY ENDPOINTS

### **Primary Endpoint**

• The change in The International Parkinson and Movement Disorder Society Nonmotor Rating Scale (MDS-NMS) (Chaudhuri 2020) total score.

**Secondary endpoints** will include changes to the following scores:

- The combined measure of The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale: Parts I, II and III(Makkos, Kovacs et al. 2018)
- The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale Part II: Motor Aspects of Experiences of Daily Living (MDS-UPDRS II) (Goetz, Tilley et al. 2008)
- The Overall Clinical Global Impressions Scale- Improvement (CGI-I) (Busner and Targum 2007)
- The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale Part III: Motor Examination (MDS-UPDRS III) (Goetz, Tilley et al. 2008)
- the Parkinson's Disease Questionnaire 39 summary index score (PDQ-39SI) (Jenkinson, Fitzpatrick et al. 1997)

## Safety endpoints

• Adverse events (AEs) frequency

• The change in the Mini Balance Evaluation Systems Test (mini-BESTest) total score (Bloem, Marinus et al. 2016)

## **Exploratory endpoints**

- The change in the following measures:
  - The Montreal Cognitive Assessment (MoCA)
  - The orally administered Symbol Digit Modality Test (oSDMT)
  - The Modified Schwab and England Activities of Daily Living Scale (S&E)
  - The Parkinson's Sleep Scale-2 (PDSS-2)
  - The Epworth Sleepiness Scale (ESS)
  - The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F)
  - The Geriatric Depression Scale (GDS)
  - The Parkinson's Anxiety Scale (PAS)
  - The Patient Reported Outcomes in Parkinson's Disease (PRO-PD)
  - The MDS-NMS Non-Motor Fluctuations (NMF) Total Score
  - The Hoehn & Yahr score (H&Y)
  - Zarit Burden Interview (ZBI)
  - Unified Parkinson's Disease Rating Scale Part I: Mentation, Behavior and Mood (UPDRS I)
  - Unified Parkinson's Disease Rating Scale Part IV: Complications of Therapy
  - EncephaLog<sup>TM</sup> Finger Tapping Test (number of finger taps)
  - EncephaLog<sup>TM</sup> Timed Up and Go Test (TUG)
    - 3-meter TUG (time to complete)
    - 10-meter TUG (stride length, cadence, rotation time, time to complete)
  - The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I: Non-Motor Aspects of Experiences of Daily Living (MDS-UPDRS I)
  - Domains of the MDS-NMS
    - Depression
    - Anxiety
    - Apathy
    - Psychosis
    - Impulse control and related disorders
    - Cognition
    - Orthostatic hypotension
    - Urinary
    - Sexual
    - Gastrointestinal
    - Sleep and wakefulness
    - Pain
    - Other

Treatment adherence and itemized answers from the following will be reported descriptively:

- a TNM<sup>TM</sup> Device usability survey
- Unified Parkinson's Disease Rating Scale Part IV (UPDRS IV)

## 3. RANDOMIZATION AND BLINDING

Upon completion of all screening and baseline assessments and verification of the inclusion and exclusion criteria, eligible study participants will be randomized on Day 29 in a 1:1 ratio using block-four randomization, stratified by site, to either the active-treatment or passive treatment condition. Additional details related to randomization can be found in section 6.3 of the STEM-PD Clinical Protocol. The active treatment will be tvCVS. In the passive treatment condition, no power will be delivered to the heating and cooling elements within the headset. However, a small amount of caloric vestibular stimulation will be transmitted upon placement of the aluminum earpieces, which will be initially cool (i.e., at room temperature) at the start of the treatment and will gradually warm to body temperature upon insertion into the participants treatment provides minimal external ear canals. This passive amount of passive stimulation that the device feasibly allows, to maintain consistency with the active treatment device. All other sensory experiences associated with device treatment will be the following: auditory tones same and include the indicating the start treatment, a faint whirring noise elicited by the cooling fans within the headset, pressure sensations felt when wearing the headset and the visual displays on the LED screen. Additionally, the choreography of starting, running and stopping a treatment will be identical for both active and passive stimulation conditions. Randomization will occur at the local site level.

## 4. SAMPLE SIZE DETERMINATION

The sample size for this study was set to achieve ~ 90% power to detect a minimal clinically important difference (MCID) of -2.64 points in the MDS-UPDRS: Part I (Horvath, Aschermann et al. 2017) for both the RCT and the first treatment period during the OLE. This estimated group sample sizes of 83 and 83 (166 total) to complete the RCT (assuming 10% attrition) achieves 89.2% power to detect a difference of 2.64 points in the MDS-UPDRS Part I total score for the null hypothesis that both group average change scores are equal and the alternative hypothesis that the average change score of the active treatment group represents greater symptomatic improvement than that of the passive treatment group given an estimated within group standard deviation of 5.32 points and a 2-sided significance level (alpha) of 0.05.

This sample size also achieves > 90% power to evaluate the primary endpoint of the STEM-PD OLE (see the STEM-PD OLE SAP for additional details).

Note that the primary outcome measure for the STEM-PD RCT is the MDS-NMS, not the MDS-UPDRS: Part I. However, the two scales are highly correlated (correlation coefficients = 0.75-0.85) (Chaudhuri, Schrag et al. 2019, van Wamelen, Martinez-Martin et al. 2021), and the MDS-UPDRS Part I has a pre-established MCID whereas the MDS-NMS does not. Given the high correlation reported for these two outcome measures in previous studies, an analysis was performed to estimate the MCID for the MDS-NMS. The MCID for the MDS-UPDRS: Part I is

2.64 points (Horvath, Aschermann et al. 2017). Since the estimated standard deviation of the MDS-UPDRS Part I for this study is 5.32 points, the MCID represents 49.6% of the standard deviation.

The standard deviation of the MDS-NMS scale has been reported as 65.87 points (Chaudhuri 2020). Using the same proportion of the standard deviation, the estimated MCID for the MDS-NMS scale for this study would be 32.7 points. Additionally, in an unpublished study analysis of participants from the original validation study, Martinez-Martin determined that among a cohort with MDS-UPDRS Part I scores greater than 10, which approximates the inclusion criterion for this study, the standard deviation of the MDS-NMS was 70.8 points. Utilizing a definition of 49.6% of the standard deviation, based upon the Martinez-Martin study, the MCID for the MDS-NMS scale would be 35.1 points.

Further, Norman et. al., 2003 (Norman, Sloan et al. 2003) suggested that the MCID be defined as 50% of the standard deviation. Using the standard deviation of 65.87, the MDS-NMS MCID would be 32.9 points. As noted above, however, the proposed study requires subjects to have an MDS-UPDRS Part I score of at least 9 at the study screen. Therefore, utilizing the standard deviation of 70.8 points (Martinez-Martin, *unpublished*), the MDS-NMS MCID would be 35.4 points<sup>2</sup>. As such, the estimated MCID range for improvement in the MDS-NMS for this Statistical Analysis Plan is -32.7 to -35.4 points. While these values provide estimates for sample size calculations, the MCID for the MDS-NMS from data collected within this study using methodology described in section 7.6.1.3.

Notably, the sample size (184 to randomize), derived from the MDS-UPDRS Part I also achieves 85.7% power to detect the estimated MCID minimum of -32.7 and 92.8% power to detect the estimated MCID maximum of -35 points in the MDS-NMS.

Competitive enrollment will be used. Participants will continue to be enrolled until at least 184 are randomized in the RCT, and if there are additional participant withdrawals, they will not be replaced. Any participant who had entered the baseline period but had not yet randomized when the competitive enrollment target is achieved may be withdrawn from the study prior to randomization, and as a result, will not be included in any of the analyses. Data from all randomized study participants will be evaluated for analyses of safety and efficacy. The protocol has planned for up to 290 study participants to be screened. The sample size of 184 to randomize allows for attrition of 10% in the RCT as well as attrition of 10% in the first treatment period of the OLE while still maintaining adequate power to evaluate the primary endpoints of those studies.

## 5. NON-COMPARATIVE INTERIM ANALYSIS

The RCT and the OLE have been designed as two portions of a single protocol with separate informed consents. This design will allow for closeout of the RCT and analysis of study data while the OLE is ongoing. However, it is possible that non-comparative, blinded interim analyses may be needed to support the Sponsor's activities, while the RCT is ongoing. As such, non-comparative analyses may be performed to evaluate the percent change in the coefficient of variation between

<sup>&</sup>lt;sup>2</sup> Protocol version 5.0 expanded eligibility criterion by lowering the MDS-UPDRS Part I threshold to 9 or more. Given this change, the standard deviation of the MDS-NMS for the total sample is estimated to be lower than 70.8 points calculated for participants with MDS-UPDRS Part I scores of 10 or more.

baseline and post treatment for the primary and secondary outcome measures using the full study cohort (i.e., pooled data from both active and passive treatment arms; allocation to remain blinded) that have both baseline and end of treatment data available. This metric provides a measure of confidence that statistical significance for a given endpoint will be achieved. This metric would be used for the purpose of fundraising. If interim analyses are performed, the results will be shared with the Independent Medical Monitor (IMM; see section 6) and Safety Medical Monitor, but results will not be shared with study site staff, investigators or Sponsor (Scion NeuroStim) staff directly involved in the trial. Results suggesting futility may be taken into consideration in the IMM recommendation to proceed or pause the study, but results indicating high probability for efficacy will not be considered as an early stopping criterion for the study. Because this noncomparative interim analysis, if performed, will be non-comparative with blinding of data unequivocally maintained and the results will not be shared with individuals who can influence the outcome of the study, the results do not pose any difficulty in terms of Type I error control or bias (Administration\_CDRH 2016). Therefore, no adjustments will be made to the alpha level for evaluating the primary or secondary endpoints using this non-comparative approach.

The interim analysis utilizes as its metric the ratio of the sample standard deviation divided by the sample mean. This metric is calculated at baseline and post treatment. The difference between these two values is divided by its baseline value as depicted in the following formula:



where:

 $\%\Delta_{SD/X}$  = the percent change in the coefficient of variation in the outcome (e.g., MDS-NMS total) score between baseline and post treatment which may be interpreted as the percent confidence that statistical significance of the outcome will be achieved in the study

 $X_{baseline}$  = the mean of the outcome scores at baseline – for outcomes collected at both baseline visits, the  $X_{baseline}$  will be the mean of the study participants' baseline scores,  $BL_{ave}$ 

 $SD_{baseline}$  = the standard deviation of the outcome scores at baseline – for outcomes collected at both baseline visits, the  $SD_{baseline}$  will be the standard deviation of the study participants'  $BL_{ave}$  scores

 $X_{post}$  = the mean of the outcome scores at the end of the treatment period  $SD_{post}$  = the standard deviation of the outcome scores at the end of treatment

For each noncomparative interim analysis, two cohorts may be evaluated. The first will be the cohort for which end of treatment data exist (i.e., data collected at either the end of the scheduled treatment period or an early termination visit). The second cohort will only evaluate data from participants that completed the visit at the end of the regularly scheduled treatment period and will exclude those with early termination from the study.

The figure below provides sample sizes that would be required to obtain percent confidence of meeting the primary endpoint assuming a change in the standard deviation of scores divided by the mean metric between the baseline and the end of treatment assessment.



Figure 1. Estimated percent confidence of achieving statistical significance in the primary endpoint according to pooled interim data collected from both treatment arms. Sample sizes that would be required to obtain percent confidence of meeting the primary endpoint assuming a change in the standard deviation of scores divided by the mean. For example, if a difference of 10% of the SD/x metric is observed in a sample of 50 participants, the metric would provide 80% confidence that the endpoint will be statistically significant at the end of the study.

## 6. INDEPENDENT DATA MONITORING

The TNM<sup>TM</sup> Device has been designated as a Non-Significant Risk Device for this study. However, the Sponsor has chosen to implement an IMM for the trial to provide independent safety monitoring and to confirm data integrity. The IMM is a physician with extensive experience in Parkinson's disease and clinical trials and has no perceived or real conflict of interest with the Sponsor or in the study outcomes. The IMM will review the research protocol and ongoing study activities with emphasis on data integrity, protocol adherence and study participant safety issues while making recommendations to the continuation, modification or conclusion of the trial. The IMM will review data at least four times per year during the course of the trial.

In addition to the IMM, the Sponsor will ensure critical safety and data points will be monitored per the STEM-PD Clinical Monitoring Plan (CMP) and the STEM-PD Data and Safety Management Plan (DSMP). A summary of key monitoring procedures is noted below:

Each site will be assigned a Clinical Research Associate (CRA) who will monitor the data to ensure the protection of rights and safety of human subjects, to verify the reported trial data are accurate, complete, and verifiable from source documents, and that the trial is conducted in compliance with the currently approved protocol/amendment(s), with Good Clinical Practice and with the applicable regulatory requirements. For all enrolled study participants, 100% source data review (SDR) and source data verification (SDV), where applicable, will occur of informed consent documents and process, demographics, inclusion and exclusion criteria, primary endpoint and key secondary endpoints (e.g., MDS-UPDRS Part III and CGI-I), all protocol deviations and safety reports, including adverse events and safety endpoints. Targeted source data verification, based on risk-based monitoring, will occur for all other endpoints and clinical data collected per the Targeted Source Data Verification (TSDV) portion of the CMP. Review of study-wide trends and key risk indicators (KRI) metrics will be reviewed in a departmental meeting to occur at least once a month. If trends are identified, the Sponsor will review with the study-assigned medical monitor and may implement a Correction and Preventative Action (CAPA) Plan, as necessary. The studyspecific Medical and Safety monitor, who has extensive experience with the device, will review and sign off on all AEs at least monthly, and all Unanticipated Adverse Device Effects (UADE) within 2 days of acknowledgment of the event. All UADEs will be reported to the ethics committees and all site Investigators per the protocol and regulatory requirements.

Previous studies with the Device have not reported any Serious Adverse Device Effects (SADEs) or UADEs. As none are anticipated for this study, if two or more serious and related adverse events (SADE or UADE) are reported, the study enrollment will pause while universality and unblinded review occurs by the Medical and Safety monitor. Additionally, the IMM will review these events for adjudication and agreement and will provide recommendations to the Sponsor.

## 7. STATISTICAL METHODS

## 7.1. GENERAL METHODS

Descriptive statistical methods will be used to summarize the data from this study, with formal hypothesis testing performed for the primary and key secondary efficacy endpoints. Unless stated otherwise, the term "descriptive statistics" refers to number of subjects, mean, median, standard deviation, minimum, and maximum for continuous data, and frequencies and percentages for categorical data. For categorical variables, the denominator of percentages will be the number of subjects in the treatment group, except for those collected by study visit and/or scheduled time point, in which case the denominator of percentages will be the number of subjects with a non-missing value at the visit and/or the scheduled time point.

All data collected during the study will be included in data listings. Unless otherwise noted, the data will be sorted first by treatment group, subject number, and then by date within each subject number.

All statistical testing will be two-sided and will be performed using a significance (alpha) level of 0.05 unless otherwise specified. P-values will be presented to three decimal places. For exploratory endpoints, inferential analyses including 95% confidence intervals and p-values will be provided, and no statements about statistical significance will be made. The p-values will be provided as informational only.

The statistical analyses will be conducted with the SAS® software package version 9.4 or higher. All analyses will be subject to formal verification procedures. Outputs will be reviewed by the lead statistician to ensure accuracy and consistency of analyses.

### 7.2. ANALYSIS POPULATIONS

**Intent-to-treat Population (ITT):** All randomized participants will be included in this population. This is the population that will be used for the primary analysis of efficacy and safety.

Modified Intent to treat (mITT): All eligible randomized participants who have completed at least one treatment with the study device and have completed a post-randomization assessment will be included in the mITT population. This population will be used for a secondary analysis of the primary endpoint and will be used to supplement the findings of the primary analysis.

**Per-protocol Population (PP):** All eligible randomized participants who (1) demonstrate at least 70% adherence of the randomized expected treatments with the Study Device<sup>3</sup>, (2) have completed the regularly scheduled end of treatment visit (day 113) (3) have not had changes to medications used to treat motor and/or non-motor symptoms of PD during the baseline or

<sup>&</sup>lt;sup>3</sup> Treatment data including dates and treatment durations are captured by the study device. These data files will be analyzed, and treatments lasting a minimum of 10 minutes will be considered as adherent for a given run based on flow oscillations in the Gossling Pulsatility Index after ~7 minutes of treatment Black, R., Rogers, L., Nicoletto, H., Adkins, H., Laskowitz, D. (2016). "Non-invasive neuromodulation using time-varying caloric vestibular stimulation - abstract." Headache 56(S1)..
RCT, (4) have not had changes to medications that mimic motor and/or non-motor symptoms of PD during the baseline or RCT will be included in the PP population. This population will be used for a secondary analysis of the primary endpoint and will be used to supplement the findings of the primary analysis and key secondary analyses.

#### 7.3. DEFINITIONS

**Study day:** The study day will be calculated in reference to the date of the first baseline virtual visit (Day 0) of the study.

**Baseline value:** Where multiple data points are collected during the baseline period, the baseline value for each participant will be calculated as the mean of assessments taken during the baseline period excluding the screening value unless otherwise noted. Exceptions to this will be for the following outcomes:

- PRO-PD where the baseline value is defined as the second data collection (i.e., first data collection will be discarded), if both are available, otherwise the first data point will be used (this value could be the Screening value). The scale's author indicated that scores from the first completion of the assessment have higher variability relative to the scores from subsequent administrations.
- the MDS-UPDRS III where the baseline value is defined as the second data collection (i.e., the in-clinic assessment). However, if the end of treatment visit is collected virtually due to the inability of the participant to attend the in-clinic visit, the data from the first virtual baseline assessment, appropriately prorated, will serve as the baseline for that participant.

To be considered baseline data, data must be collected prior to or on the day of first treatment with the study Device.

**Duration of Follow-up:** The duration of follow-up will be defined as the number of days from Baseline Visit 1 until the End of Study assessment or the last completed visit (phone call, virtual or in clinic).

#### **Adverse Event:**

Per protocol, an AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, users, or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device and the events related to the procedures involved. For purposes of analyses, any AE specified on the Adverse Events eCRF page is considered an AE.

#### **Adverse Device Effect (ADE):**

Per protocol, an ADE is an AE related to the use of an investigational medical device. For purposes of analysis, any AE specified on the Adverse Events eCRF page that is possibly related, probably related, or related to the study device will be considered an ADE.

#### **Serious Adverse Event (SAE):**

Per protocol, a SAE is an AE that has

- Led to death,
- Led to serious deterioration in the health of the participant, that either resulted in:
  - 1. A life-threatening illness or injury, or
  - 2. A permanent impairment of a body structure or a body function, or
  - 3. In-patient or prolonged hospitalization, or
  - 4. Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or body function.
- Led to fetal distress, fetal death or congenital abnormality or birth defect.

For analysis purposes, SAEs are AEs which are defined as serious on the Adverse Events eCRF (page 103).

## **Serious Adverse Device Effect (SADE):**

Per protocol, a SADE is an ADE that has resulted in any of the consequences characteristic of a serious adverse event. For analysis purposes, any AE on the Adverse Events eCRF page that is possibly related, probably related, or related to the study device and is noted as serious will be considered a SADE.

#### **Unexpected Adverse Device Effect (UADE):**

Per protocol, a UADE is an SADE on health or safety or any life-threatening problem or death caused by, or associated with, a device, if that effect problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of participants. For analysis purposes, any event noted on the SADE/UADE Report eCRF page that is noted as a UADE will be considered a UADE.

SADEs and UADEs are AEs specified as such on page 111 of the eCRF. More information on SAEs, ADEs, SADEs, and UADEs can be found in Protocol (Version 6.0: 02 Apr 2024) Section 8.2.

## 7.4. ANALYSIS OF STUDY CONDUCT

The number of participants screened and the number of those randomized falling into the ITT, mITT and PP populations will be summarized.

Study treatment administration, duration of follow-up, discontinuation from study treatment and the reasons for discontinuation will be summarized by treatment group for all randomized participants. Coded protocol deviations and protocol violations will also be summarized as follows:

• Major/Important versus Minor versus No Impact, where:

- Major/Important are protocol deviations that might significantly impact completeness, accuracy, and/or reliability of study data OR could significantly affect a participant's rights, safety or well-being
- Minor are protocol deviations with minor impact on data quality or patient safety
- No impact are protocol deviations that do not impact data quality or patient safety
- Specific subcategories of coded deviations and violations will be further summarized by treatment group.

#### 7.5. DESCRIPTION OF THE DATASET USED FOR ANALYSIS

SAS-compatible data sets will be exported directly from the iMediData RAVE Electronic Data Capture platform. Exceptions may include data for the MDS-UPDRS Part III that has been scored by central blinded raters within the Machine Medicine Kelvin-PD platform, data related to Finger-tapping tests and Timed Up and Go tests captured with the Mon4t EncephaLog application, treatment adherence data downloaded from the returned study Devices, a file that defines types of medications taken to address motor and nonmotor symptoms of PD including the levodopa equivalent daily dose for each randomized participant, the list of centers that required inclusion of the Sponsor name on the informed consent forms, and a file that defines all the assignment of each consented participant into populations for analysis (e.g., ITT, mITT and PP) and reasons for exclusion and withdrawal where appropriate. Data for these exceptions will be provided as csv files created with Microsoft Excel.

#### 7.6. ANALYSIS OF TREATMENT GROUP COMPARABILITY

An evaluation of treatment group characteristics will be compared across the two treatment arms. The characteristics will include demographics, baseline disease characteristics, concomitant medications, scores in outcome measures at baseline. Descriptive statistics will be presented by treatment groups. Differences in baseline scores will be determined using parametric or non-parametric approaches as appropriate based upon visual inspection of the distribution. Categorical variables will be summarized using frequencies and percentages. Baselines will be considered different in circumstances where p < 0.05. Numbers of early withdrawals will be compared across treatment arms using Fisher's exact test. Reasons provided for early post-randomization withdrawals will be reported. Withdrawals due to similar adverse events will be grouped into categories. Fisher's exact tests stratified by category will then be conducted to determine if there is an association between the number of subjects experiencing withdrawal due to adverse events and treatment arm.

#### 7.6.1. Demographics and Baseline Characteristics

The following characteristics will be summarized for participants in each treatment group and each cohort (i.e., ITT, mITT and PP): age, sex, years since PD diagnosis, levodopa equivalent daily dose (LEDD) at start of treatment (Jost, Kaldenbach et al. 2023), race and ethnicity.

#### 7.6.2. Disease characteristics

Baseline Hoehn & Yahr scores will be summarized. Additionally, motor phenotypes (i.e., tremor-dominant, postural instability gait difficulty and intermediate) classified based on the Baseline 2 visit MDS-UPDRS part II and part III scores and previously-established methodology (Stebbins, Goetz et al. 2013). Specifically, a Tremor score will be calculated by summing all items from 2.10, 3.15, 3.16, 3.17 and 3.18 from the MDS-UPDRS. A postural instability and gait difficulty (PIGD) score will be calculated by summing all items from 2.12, 2.13, 3.10, 3.11 and 3.12 from the MDS-UPDRS. Ratios of Tremor score/PIGD score will be used to classify motor phenotypes. Ratios ≥1.15 = Tremor dominant. Ratios ≤0.90 = PIGD dominant. Scores > 0.9 and <1.15 = intermediate. If data required to calculate the scores is missing from the Baseline 2 visit, data from the Baseline 1 visit will be analyzed. Post randomization data will not be considered. Classification will only be performed on complete case data.

#### 7.6.3. Pre-study and Concomitant Medications

The number and percentage of each treatment group on concomitant therapies at randomization will be reported categorically including the following:

- adenosine A2A antagonists
- amantadine
- anticonvulsants
- anti-depressant/antianxiety medications
- antiemetics
- antihistamines
- antihypertensives
- antipsychotics
- central anticholinergies
- cognitive enhancers
- COMT Inhibitors
- contraceptives
- corticosteroids
- dystonia treatments
- incontinence treatments
- inhaled levodopa
- inhaled or ingested cannabinoids
- laxatives/stool softeners
- MAO-B inhibitors
- narcotics
- oral or transdermal dopamine agonists
- oral levodopa-based therapies
- oral levodopa-based therapies/COMT inhibitors
- orthostatic hypotension treatments

- pain/cramping treatments
- pump therapies
- sexual dysfunction treatments
- sialorrhea treatments
- sleep aids
- stimulants
- other

Changes in medications to treat symptoms associated with PD during the trial are a protocol deviation. Changes in these medications would exclude participants from the PP analysis and will be determined prior to unblinding of treatment allocation. Changes in medications used to treat symptoms associated with PD and change from baseline to end of treatment in LEDD will be summarized descriptively for the mITT and the ITT populations.

Certain concomitant medications (e.g., antihistamines, central anticholinergics or acetylcholinesterase inhibitors) may alter treatment efficacy by affecting neurotransmitter systems involved in the mechanisms of action for tvCVS. Sensitivity analyses will be performed to compare treatment effects in study participants taking these concomitant medications during the trial against study participants that did not take these concomitant medications.

## 7.6.4. Study Device Administration

Treatment adherence will be analyzed after the database lock for the RCT. Treatment adherence data will be reported descriptively. Treatment adherence  $\geq 70\%$  of the expected randomized treatments over the duration of the treatment period will be required for inclusion in the PP analysis (see section 7.1).

#### 7.7. EFFICACY ANALYSIS

Efficacy will be determined using (Zeger and Liang 1992, Zorn 2001) a linear regression utilizing a mixed effects (i.e., mixed model repeated measures [MMRM]). This approach allows for repeated measurements on a subject (i.e., all time points during the study) and unequally spaced as well as missing data (dropouts or intermittent), allows for the inclusion of continuous or categorical covariates, allows for a flexible specification of the covariance structure. This modeling technique has been shown to produce unbiased estimates in the case of data missing at random. Additionally, the MMRM estimation is robust to departures from normality. (Rubin 1987)

The following MMRM model (Zeger and Liang 1992, Zorn 2001) will be analyzed to determine significance for the primary endpoint:

$$\begin{split} Y_{ij} \sim N(0, &\sigma^2) \\ Y_{ij} = \beta_0 + \beta_1 * ARM_i + \beta_2 * VISIT_{ij} + \beta_3 * ARM_i * VISIT_{ij} + \beta_4 * SITE_i \\ where: \end{split}$$

 $Y_{ij} = (MDS\_NMS \text{ total score for participant i at time j}) - (MDS\_NMS \text{ total score for } j)$ 

participant i at baseline),

 $ARM_i = 1$  if participant i is in the treatment arm

= 0 if participant i is in the passive arm,

 $VISIT_{ij}$  = an ordinal variable representing the visit for  $j^{th}$  measurement for participant i

SITE<sub>i</sub> is a nominal variable indicating the site for participant i,

An unstructured covariance structure will be utilized for the R matrix. The Kenward-Roger approximation will be used to estimate the denominator degrees of freedom. The difference between active and passive treatment at each visit will be estimated based on the Least Squares Mean (LSMean) difference between the treatment groups at the visit from the MMRM with the associated 90% confidence interval (CI) and 1-sided P-value. Additionally, the p-value for the site effect will be presented. If the unstructured covariance matrix results in convergence issue, the heterogeneous Toeplitz covariance structure followed by the heterogeneous first-order autoregressive (AR(1)) structure will be used. In these cases, sandwich estimators will be obtained from the model fitting procedure to ensure unbiased estimation of the treatment effect.

Note: The VISIT effect will be included only when there are multiple post-randomization assessments for a given endpoint. In those cases, a significant interaction between ARM and VISIT will determine a statistically significant finding at a given VISIT. An effect for baseline value will be included for outcomes where the baseline scores significantly different between the treatment arms.

In cases where there is a single post-randomization assessment for a given endpoint, the linear model fit will be simplified to:

```
\begin{split} Y_i &\sim N(0, \sigma^2) \\ Y_i &= \beta_0 + \beta_1 * ARM_i \ + \beta_2 * SITE_i \\ \text{where:} \\ Y_i &= (\text{Endpoint assessment for subject i}) - (\text{Endpoint assessment for participant i at baseline}), \\ ARM_i &= 1 \text{ if participant i is in the treatment arm} \\ &= 0 \text{ if participant i is in the passive arm,} \end{split}
```

SITE<sub>i</sub> is a nominal variable indicating the site for participant i,

The difference between active and passive treatment will be estimated based on the Least Squares Mean (LSMean) difference between the treatment groups from the linear model with the associated confidence interval (CI) and P-value. Additionally, the p-value for the site effect will be presented.

An effect for baseline value will be included for outcomes where the baseline scores significantly different between the treatment arms.

## 7.7.1. Primary Endpoint

The primary endpoint is the change in MDS-NMS total score at the end of the treatment period (day 113) relative to baseline (mean of day 0 and day 29) scores.

## 7.7.1.1. Statistical Significance

The null hypothesis is TNM<sup>TM</sup> Device treatments will yield an equivalent change in NMS burden in the two treatment arms. The alternative hypothesis is that the active treatment arm will do better than (be superior to) the passive treatment arm. The threshold to determine statistical significance will be set at  $\alpha = 0.05$  based upon a 1-tailed test<sup>4</sup>.

## 7.7.1.2. Clinical Significance

Clinical significance is determined by how a treatment affects the extent to which a participant is currently living independent of help from others OR that there is a real genuine, palpable, and noticeable effect on daily life or how a patient feels, functions, or survives. Importantly, as the scores from the MDS-NMS are derived from the product of the symptom frequency (how often the participant has experienced a given non-motor symptom since the last evaluation with higher scores indicating more frequent experience) and the symptom severity (impact of that symptom on how the participant has felt and functioned with higher scores indicating greater distress or disturbance to patient or caregiver), reductions in MDS-NMS total scores are inherently clinically meaningful in that they represent how the participant is feeling and functioning. Given the inherent clinical meaningfulness of the MDS-NMS total score, the primary endpoint will be considered clinically meaningful, and therefore, successful, if there is a statistically significant reduction in MDS-NMS total scores in the active tvCVS group relative to the passive treatment group after 12 weeks of twice-daily treatment.

## 7.7.1.3. Supportive analysis to further explore clinical significance

The structure and methodology for data collection of the MDS-NMS allows for statistically significant changes to be interpreted as inherently clinically meaningful. However, the scale is relatively new and may not be well known by all prescribing/referring physicians. Therefore, to facilitate clinical adoption, a supplementary analysis will be performed that establishes a minimal clinically important difference (MCID) for the MDS-NMS within the study. The MCID will be defined using an anchor-based approach and will be defined as the average of the

<sup>&</sup>lt;sup>4</sup> Regulatory review within certain bodies (e.g., the United Kingdom) may require that the endpoint results meet a threshold with an alpha of 0.025 based upon a 1-tailed test. Therefore, this higher level of significance will also be evaluated for certain premarket submissions.

MCIDs estimated from a compilation of data from both the intervention (active treatment) and the control (passive treatment) arms for two distinct anchors.

These anchors include (1) the Non-Motor Symptom-focused Clinical Global Impressions Scale – Improvement (NMS CGI-I), part of the Focused CGI-I, and (2) the Non-Motor Symptom Burden transition question (Transition Questionnaire). The NMS CGI-I is a clinician-rated scale that is based on account information gathered through interviews with the study participant and the study partner and through the review of medical records. The NMS CGI-I will evaluate clinically meaningful change between the baseline and the end of the treatment period. The Non-Motor Symptom Burden question (Transition Questionnaire) will capture participant reports of perceived change in overall NMS burden after four weeks of treatment compared to the period before starting treatment with the device.

These two anchors will be collected at the same study visits or on the ePRO data collection associated with the MDS-NMS data collection on Treatment Visit 1 (day 57). This data collection will allow for sufficient power to calculate the receiver operating characteristic curve (ROC) with 95% confidence and 80% Power (Figure 2). Spearman correlation coefficients will then be calculated to determine, separately, the relationship between each of these measures and changes in the MDS-NMS score. Assuming that both measures show correlation coefficient with magnitude of at least 0.5, the following steps will be undertaken. ROC curves will be developed separately the measures to determine cutoff values define the MCID calculated with that anchor (Kumar and Indrayan 2011). Note that for NMS-focused CGI-I, the standard approach of utilizing ROC analysis to determine the optimal cutoff value in the MDS-NMS Total Score that best distinguishes 'minimally improved' (score of 3) from 'no change' (score of 4) (Hauser, Auinger et al. 2011, Horvath, Aschermann et al. 2015, Falissard, Sapin et al. 2016, Czobor, Sebe et al. 2022, Christensen, Adair et al. 2023) will be performed. For the Non-Motor Symptom Burden transition question (Transition Questionnaire), the ROC will be developed to calculate the cutoff value in the MDS-NMS Total Score that best distinguishes 'mildly better' from 'no change'. For each measure, because the risks of false positive and false negative may not be equal, Youden's J statistic will be used to determine the MCID (Youden 1950)

$$J = \frac{ad - bc}{(a+b)(c+d)}$$

and a, b, c, and d are subject counts defined from:

| | | Based on | Measure |
|------------------|---------------|-----------|---------------|
| | | Improving | Not improving |
| Decedes Analysis | Improving | а | b |
| Based on Anchor | Not Improving | С | d |

The largest J statistic value for both ROC curves will define the MCIDs for each of the two anchors (i.e., the NMS CGI-I and the Non-Motor Symptom Burden transition questionnaire).

Having now obtained two separate estimates for the MCID, the weighted average, where the correlation squared (r<sup>2</sup>) value will be the associated weight, will then be utilized to determine the operationalized MCID. If exactly one of the two Spearman correlation coefficients previously calculated to determine relationships between each measure and the change in the MDS-NMS score has a magnitude below 0.5, then that measure will be disregarded, and the MCID will be determined solely for the measure that had correlation coefficient of at least 0.5. Lastly, if both of the Spearman correlation coefficients have magnitudes below 0.5, then a distribution-based approach will be utilized to determine the MCID. The distribution-based method would be performed wherein the distribution of MDS-NMS Total Scores at baseline are used to determine the standard deviation of the baseline scores. This value is then multiplied by 0.3 to determine the MCID as 0.3 is defined as a small effect size (Anderson, Kelley et al. 2017). To support the conclusions of this distribution-based method of defining the MCID, a correlation analysis evaluating changes in the MDS-NMS and the MDS-UPDRS Part I may also be conducted as the latter is known to strongly correlate with the MDS-NMS and has a previously established MCID of 2.64 points (Horvath, Aschermann et al. 2017).



**Figure 2: Sample size requirements for ROC curve analysis**. Note: It is expected that the area under the ROC curve (AUC) will have a value between 0.65 and 0.75.

Once the MCID is determined, it can be used to calculate the percentage of cases that exceed that value for each of the two treatment arms (i.e., responder rates). To further support clinical adoption, a supporting Fisher's exact test analysis will be employed to determine if the responder rate for active treatment participants is statistically significantly greater than the response rate for passive treatment participants. For statistical significance, the required percentage of participants in the intervention group that demonstrate a change exceeding the MCID will be a function of the percentage of participants in the passive treatment group that demonstrate a change exceeding the MCID. This relationship is depicted in Figure 3. Because the power of this binomial comparison will be reduced under conditions where there is a high rate of passive treatment participants that exceed the MCID, if 36% or more of the passive treatment arm exceeds the MCID (a condition that would require > 60% responder rate in the active arm), clinical significance for the primary outcome measure will instead be further supported by verifying that the mean/median difference between the two treatment arms exceeds the change equivalent to the MCID.



Figure 3: Effect of Percent in Passive Group Exceeding MCID on the Required Percent of Active Group Needing to Exceed MCID to demonstrate statistical significance using binomial comparison.

Additional analyses of the primary endpoint measure to support clinical adoption will include the following:

• The percent change of scores (normalized to the average baseline)

The percent change of scores is calculated as the mean change score divided by the mean baseline value multiplied by 100.

• The percentage of participants who improved by 1 MCID or more (i.e., change from baseline in MDS-NMS Total Score at Day 113 ≥ MCID calculated on an individual level). Participants who do not meet this criterion are non-responders.

The proportion of participants whose change from baseline to Day 113 in NMS-MDS total score met or exceeded the MCID will be summarized by treatment group.

#### Effect Sizes

Effect size will be calculated in two ways:

- a. Cohen's w will be calculated for the 2x2 table of responders/non-responders and treatment group. Cohen's w is calculated as the square root of the chi-square test statistic divided by the total number of participants. Responders are defined as those participants with change from baseline in MDS-NMS Total Score at Day 113 ≥1 MCID. Non-responders are those who did not respond (includes missing data as non-responders).
- b. Cohen's D will be derived as the ratio of the estimated difference in the change from baseline MDS-NMS to the population standard deviation at each visit estimated from the model (the square root of the diagonal elements of the estimated covariance matrix).
- The number needed to treat to obtain 1 patient with improvement of 1 MCID or more

The number needed to treat is calculated as 1/the absolute difference between treatment groups in the proportion of non-responders (i.e., change from baseline in MDS-NMS Total Score at Day 113 < MCID or missing).

#### • Reliable Change Index

Reliable Change Index is defined per participant as the difference of the pre and post treatment scores divided by the standard error of the measurement. The standard error of the measurement is calculated as the square root of two times the standard error of the mean difference between pre and post treatment scores, squared ( $\sqrt{2(SEM^2)}$ ). This value is compared to the cutoff score assuming a normal distribution and 95% confidence level. The proportion of values above (RC+), below (RC-), and at (RCo) the cutoff value will be presented. This value will be calculated for the change from baseline in MDS-NMS Total scores at Day 113.

#### • Cumulative Distribution Plot

A plot of the cumulative distribution of the change from baseline in MDS-NMS Total scores at Day 113 will be prepared.

## 7.7.2. Secondary Endpoints

Multiplicity of study endpoints will be adjusted for using a hierarchical strategy whereby endpoints in the study are only considered to be statistically significant if both of the following are true: 1) p < 0.05 AND 2) the preceding endpoint was found to be statistically significant at the significance level  $\alpha = 0.05$ . More specifically, the hierarchical order for evaluation of efficacy endpoints is the following: MDS-NMS Total Score (primary endpoint); the combined measure of MDS-UPDRS Parts I, II and III (secondary endpoint), MDS-UPDRS part II (secondary endpoint); Overall CGI-I (secondary endpoint); MDS-UPDRS part III (secondary endpoint); PDQ-39SI (secondary endpoint). Note that all the secondary endpoints have an *a priori* direction, thus one-tailed tests will be utilized for analyses. Only participants who have baseline data collected for the secondary endpoints will be included in these efficacy analyses.

## 7.7.2.1. Combined measure of MDS-UPDRS Parts I, II, and III (sum score)

This endpoint will evaluate the change in the combined measure of MDS-UPDRS Parts I, II and III at the end of the treatment period (day 112 and 113), which is defined based on the change relative to baseline (days 28/29) scores to provide a measure of global function in PD. This outcome will support that TNM<sup>TM</sup> Device treatment provide clinically meaningful changes for people with PD. Changes meeting or exceeding the previously established MCID for this measure (-6.7 points for clinical improvement) (Makkos, Kovacs et al. 2018) will be considered clinically meaningful. MDS-UPDRS Part II.

This endpoint will evaluate the change in MDS-UPDRS part II score at the end of the treatment period (day 112) relative to baseline (mean of day 0 and day 28) scores. Changes will be considered to be clinically meaningful if the mean difference (if normal distribution) or median difference (if non-normal distribution) meets or exceeds the previously established MCID (-3.05 for clinical improvement) (Horvath, Aschermann et al. 2017).

#### 7.7.2.2. Overall CGI-I

This endpoint will evaluate the CGI-I score at the end of the treatment period (day 113) which is defined based on change relative to baseline evaluation at day 29. This CGI-I provides a clinician's determination of overall change as it relates to all aspects of PD. For ease of interpretation, the CGI-I score will be converted using the following formula: Converted CGI-I = 4 – CGI-I. Thus a 0 corresponds to no change, higher magnitude positive values correspond to greater improvements and higher magnitude negative scores correspond to increased worsening. To allow for an effect of site, treatment differences will be modeled utilizing the MMRM with no effect for visit as described previously. If the active treatment arm demonstrates converted CGI-I scores that are statistically significantly greater than those in the passive treatment arm, these results would further support the clinical meaningfulness of change due to tvCVS.

#### 7.7.2.3. MDS-UPDRS Part III

This endpoint will evaluate the change in MDS-UPDRS Part III score at the end of the treatment period (day 113) relative to the baseline (day 29) score. Changes will be considered to be clinically meaningful if the mean/median difference meets or exceeds the previously established MCID (-3.25 for clinical improvement) for this scale (Horvath, Aschermann et al. 2015).

This analysis will be derived only from the ON-state MDS-UPDRS Part III: motor exam scores, and MDS-UPDRS Part III data collected in the OFF-state will not be included in any analysis. The scores will be provided by blinded central raters when available except for scores from item 3 (related to rigidity). Scores for items related to rigidity will be derived from the blinded local rater scores when calculating the MDS-UPDRS part III score. Additionally, the ability of the centralized raters to provide scores will depend on the availability of quality video feed captured by the clinical sites. Video will be captured by Machine Medicine's Kelvin-PD software which was selected by the Sponsor to minimize the risk of video capture that is of inadequate quality for accurate centralized rating. However, it is possible that some video data may be missing or of poor quality, and thus, cannot be rated by a central rater. In cases where MDS-UPDRS Part III data from central raters from either the baseline or the end of treatment visit cannot be scored by the central rater, scores provided by the local raters will be utilized for both the baseline and end of treatment assessments. In cases where the last assessment was captured remotely using telemedicine platforms, the score will be prorated to the scale of the in-clinic MDS-UPDRS Part III. Additionally, the day 0 baseline measure (virtual visit) will be prorated to the scale of the in-clinic MDS-UPDRS Part III will be substituted for the baseline value. This will only occur if a virtual visit is required due to the participant's inability to travel to the site for the end of treatment visit.

\* Some motor examinations will be rated by multiple raters to establish inter-rater reliability and approve central raters. Analysis of efficacy should only be performed for the rater assigned by the Sponsor for a given participant or assessment. Additionally, some raters may wish to go back and re-rate an examination. In cases where one rater has performed multiple scores, the most recent score should be utilized in the analysis of efficacy and all prior ratings should be ignored.

# 7.7.2.4. PDQ-39SI

This endpoint will evaluate the change in PDQ-39SI score at the end of the treatment period (day 112) relative to baseline (mean of day 0 and day 28) scores. The PDQ-39SI is derived by the sum of the eight PDQ-39 scale scores divided by eight (the number of scales), which yields a score between 0 and 100 (with a score of 100 indicating more health problems) (Jenkinson, Fitzpatrick et al. 1997). This is equivalent to expressing the sum of all 39 item responses as a percentage score. Changes will be considered to be clinically meaningful if the mean/median difference meets or exceeds the previously

established MCID (-4.72 for clinical improvement) for this scale (Horvath, Aschermann et al. 2017).

#### 7.8. SAFETY ANALYSIS

## 7.8.1. Adverse Events (AEs)

Participants will be assessed for AEs every two weeks at minimum (either at study visits or during phone calls). For each group, the AEs will be summarized with frequency and percentage by preferred (PT) term, with all participants in that treatment group as the denominator. Classification will utilize MedDRA System Organ Class (SOC) based on MedDRA® Version 26.0 or other terminology/classification common to Parkinson's disease (e.g., falls, freezing of gait, etc.). AE incidence will be summarized by both severity and causal relationship to Device treatment (as determined by the blinded Principal Investigator or designated study personnel). AEs deemed to be of "possible" or "probable" relationship or "related" to the Device will also be considered as device related. AEs that occurred during the baseline period and post randomization will also be summarized. Additionally, the number of events and number of device-related events per person will be reported as a distribution.

The AE summary tables will provide an overall summary of AEs including the number and percentage of participants who experienced any AE, any SAE, any ADE, any SADE, any UADE, and any discontinuations in study participation due to an AE. Differences between the two arms for each AE type will be evaluated by a Fisher's exact test.

## 7.8.2. Safety Endpoint

The change in the mini-BESTest between the end of treatment (day 113 or early withdrawal) and the baseline (day 29) will serve as an additional safety endpoint to confirm that TNM<sup>TM</sup> treatment does not negatively impact balance, functional mobility and gait in people with PD. Mini-BESTest data collected in the OFF-state will not be included in any analysis. The largest amount by which the median change scores in the passive treatment arm can be better than the median change scores in the active treatment arm is 4 points (Godi, Franchignoni et al. 2013). Two-sided, 95% confidence intervals for the median difference in the Mini-BESTest scores for the two treatment groups will be constructed (Ganju and Rom 2017). If the confidence interval of the difference (active – passive) contains -4, then the no clinically meaningful difference between the groups exists.

#### 7.9. EXPLORATORY ANALYSES

These exploratory endpoints have been added to support clinical applicability of the primary and secondary endpoints. They have been selected to provide additional details that will impact decisions made by prescribing physicians and reimbursement entities. Mean or median change with corresponding 95% confidence intervals and p values will be provided. No adjustments will be made to address a multiplicity of endpoints. Only participants who have

baseline data collected for the exploratory endpoints will be included in these efficacy analyses.

Only participants who have baseline data collected for the exploratory endpoints will be included in these efficacy analyses.

- 1. The Montreal Cognitive Assessment (MoCA): This endpoint will evaluate the change in MoCA score at the end of the treatment period (day 113) relative to the baseline (day 29). The MoCA collected at the study screen will be used to evaluate study eligibility only and will not be included in the analysis.
- 2. The Oral Symbol Digit Modality Test (oSDMT): This endpoint will evaluate the change in oSDMT score (total correct substitutions) at the end of the treatment period (day 113) relative to the baseline (day 29).
- 3. The Modified Schwab and England Activities of Daily Living Scale (S&E): This endpoint will evaluate the change in S&E score at the end of the treatment period (day 113) relative to the baseline (day 29).
- 4. The Parkinson's Disease Sleep Scale-2 (PDSS-2): This endpoint will evaluate the change in PDSS-2 score at the end of the treatment period (day 112) relative to the baseline (day 28).
- 5. The Epworth Sleepiness Scale (ESS): This endpoint will evaluate the change in ESS score at the end of the treatment period (day 112) relative to the baseline (day 28).
- 6. The Functional Assessment of Chronic Illness Therapy-Fatigue Scale (FACIT-F): This endpoint will evaluate the change in FACIT-F score at the end of the treatment period (day 112) relative to the baseline (day 28).
- 7. The Geriatric Depression Scale (GDS): This endpoint will evaluate the change in GDS score at the end of the treatment period (day 112) relative to the baseline (day 28).
- 8. The Parkinson's Anxiety Scale (PAS): This endpoint will evaluate the change in PAS score at the end of the treatment period (day 112) relative to the baseline (day 28).
- 9. The Patient Reported Outcome Parkinson's Disease (PRO-PD): This endpoint will evaluate the change in the PRO-PD score at the end of the treatment period (day 113) relative to the baseline (day 29). The PRO-PD collected at the study screen will be used as a practice-only and will not be included in the analysis as the scale's author indicated that scores from the first completion of the assessment typically have high variability relative to the scores from subsequent administrations. However, in cases where the PRO-PD was collected at the study screen but not day 29 (missing data), the score at the study screen will be used for the baseline measure.
- 10. The MDS-NMS Non-Motor Fluctuations (NMF) Total Score: This endpoint will evaluate the change in NMF score at the end of the treatment period (day 113) relative to the baseline (day 29).
- 11. The Hoehn & Yahr score: This endpoint will evaluate the change in H&Y score at the end of the treatment period (day 113) relative to the baseline (day 29).
- 12. Zarit Burden Interview (ZBI): This endpoint will evaluate the change in ZBI score at the end of the treatment period (day 113) relative to the baseline (day 29).
- 13. The Unified Parkinson's Disease Rating Scale Part I (UPDRS I) This endpoint will evaluate the change in UPDRS I score at the end of the treatment period (day 113) relative to the baseline (day 29).
- 14. EncephaLog<sup>TM</sup> Finger Tapping Test This endpoint will evaluate the change in the number of total finger tap (left and right hands combined) at the end of the treatment period (day 112)

relative to the baseline (mean of data collected prior to randomization).

- 15. EncephaLog<sup>TM</sup> 3 meter Timed Up and Go Test (3m TUG) 3m TUG at home in the clinic: This endpoint will evaluate the change in the duration of the 3m TUG at the end of the treatment period (day 112) relative to the baseline (mean of data collected weekly prior to randomization).
- 16. EncephaLog<sup>TM</sup> 10 meter Timed Up and Go Test (10m TUG) This endpoint will evaluate the change in the average of replicate values taken for several measures related to the conduct of the 10m TUG at the end of the treatment period (day 113) relative to the baseline (day 29) including stride length, cadence, rotation time, time to complete.
- 17. The International Parkinson and Movement Disorder Society Unified Parkinson's Disease Rating Scale Part I: Non-Motor Aspects of Experiences of Daily Living (MDS-UPDRS I): This endpoint will evaluate the change in MDS-UPDRS I score at the end of the treatment period (day 113) relative to the baseline (day 29).

Treatment adherence,  $TNM^{TM}$ Device usability/satisfaction (Device Useability Questionnaire) and itemized answers from UPDRS IV assessment tool will also be reported descriptively. To further explore the effects of treatment on individual NMS, effects of treatment on each of the individual MDS-NMS domains will be evaluated. These domains include the following: (1) Depression, (2) Anxiety, (3) Apathy, (4) Psychosis, (5) Impulse control and related disorders, (6) Cognition, (7) Orthostatic hypotension, (8) Urinary, (9) Sexual, (10) Gastrointestinal, (11) Sleep and wakefulness, (12) Pain, and (13) Other. As this is an exploratory analysis, as opposed to a primary or secondary aim, only subjects that demonstrate burden in the specified domain will be evaluated. In practice, this means that if any subject shows no burden on a given MDS-NMS domain throughout the study, then they will be excluded from this exploratory analysis.

#### 7.10. ADDITIONAL SENSITIVITY ANALYSES

#### 7.10.1. Item-level Missing Data

For MDS-NMS and MDS-UPDRS Parts I, II, and III, missing item-level scores may be imputed under certain circumstances. For MDS-NMS, a missing item-level score may be imputed with the average of the non-missing items for a given domain provided that there is no more than 40% missingness within that domain. This means that missing items from a 2-question domain may not be imputed. If all items in a domain are not scored after the item level imputation, that domain score is considered as missing, and the corresponding total score will be missing.

For MDS-UPDRS Part I, a single item-level missing value can be imputed with the average of the non-missing values for that Part if no more than 1 missing values exists. For MDS-UPDRS Part II, item-level missing values can be imputed with the average of the non-missing values for that Part if no more than 2 missing values exist. For MDS-UPDRS Part III (in-clinic assessment), item-level missing values can be imputed with the average of the non-missing values for that Part if no more than 7 missing values (Goetz, Luo et al. 2015).

For MDS-UPDRS Part III captured virtually and MDS-UPDRS Part IV, no item level missing values will be imputed.

# 7.10.2. Missing data

The study protocol has been designed with the objective of minimizing missing data as much as possible. The Study Device has been designated as a Non-Significant Risk Device by the US FDA. Furthermore, the same treatment waveforms that will be used in this study were found to be highly tolerable in previous studies in PD (Wilkinson, Podlewska et al. 2016, Wilkinson, Podlewska et al. 2019, Wilkinson, Podlewska et al. 2019) and episodic migraine (Wilkinson, Ade et al. 2017). Therefore, it is anticipated that any data missing in this trial will be at random and not a result of the treatment arm. Analysis will be conducted using MMRM to allow for unbiased estimation of treatment effect in the presence of missingness at random. (Yuan 2014)For the full MDS-UPDRS Part III collected at the baseline visit 2 (day 29) and end of treatment visit (113) and not collected during baseline 1 (day 0) and interim visits at days 57 and 85, missing item-level values will be imputed using the method described in the previous section. If a missing Day 113 assessment exists after the item level imputation, then the last available post-baseline virtual assessment (Day 57 or Day 85) will be imputed after the value has been prorated using the formula: prorated value = virtual value\*(132/108). If this value is utilized the suitably prorated value for Baseline 1 (Day 0) will be utilized rather than the Baseline 2 (Day 29) value. (Rashid 2021) These imputed values for missing data would be applied to both the composite measure for MDS-UPDRS I, II & III and the MDS-UPDRS III secondary outcome measures.

#### 7.10.3. Protocol Deviations

To demonstrate the robustness of confounding protocol deviations or violations that impact the interpretation of efficacy analyses, subgroup analyses will be performed utilizing the absence/presence of a confounding deviation to the that element of the protocol (i.e., a change in medication that mimics symptoms of Parkinson's disease occurred, a change in medication used to treat motor and/or non-motor symptoms of Parkinson's disease occurred and/or data was collected at a visit performed out of window when the participant was not treating when protocol requires). Subgroup analyses will be conducted for the primary outcome, the combined measure of the MDS-UPDRS Parts I, II, and III and Mini-BESTest at minimum.

#### 7.10.4. Study blind

Although unlikely, it is possible that knowledge of the study Sponsor and Device name may have the potential to unblind participants or bias them with regard to their expectation of treatment effect. Therefore, the study Sponsor excluded this information from informed consent documents. However, a subset of local institutional review boards and ethics committees required that the Sponsor name be included in the informed consent forms given to the participants at their site. To determine if having the name of the Sponsor in

the informed consent alters the effect of the device, the same modeling methodology used for the efficacy analysis described above will be utilized to determine the effect of having knowledge of the Sponsor name on efficacy, specifically, MMRM will be utilized separately for participants treated at sites where the Sponsor name was included in the ICF vs not included in the ICF. The results of this analysis will be used to determine if knowledge of the Sponsor name affects the relationship between treatment (active or passive) and each outcome. This analysis will be conducted for primary and secondary outcomes.

#### 7.10.5. Comparison to baseline 2

For the primary outcome (at minimum), a confirmatory sensitivity analysis will be conducted to evaluate change in the primary outcome relative to scores obtained during the second baseline assessment only.

# 7.10.6. Physical limitations

The mini-BESTest (a safety outcome) provides a measure of balance, functional mobility and gait. However, certain aspects of the scale may be negatively impacted due to temporary physical limitations (e.g., lower leg injury) and would be negatively impacted if data was collected in the off-state. Therefore, a confirmatory sensitivity analysis may be conducted that excludes data from study participants that either could not complete all elements of the scale due to bodily injury or impairment (as identified by the scale's rater or ongoing adverse events) or whose data was collected in an off state.

# 7.10.7. Country and Other Subgroups

An analysis of the primary endpoint and select secondary endpoints will be conducted by country to determine if there is a different treatment effect in the United Kingdom as compared to the United States. For this analysis, separate models will be constructed per subgroup.

Other primary endpoint and select secondary endpoint subgroups to be evaluated include: Sponsor name utilized in ICF (Sponsor name in ICF vs Sponsor not in ICF), Prohibited Concomitant Medication Use (Used vs Not Used), the subset of confounding protocol deviations as noted in section 7.10.3, specifically, a change in medication that mimics symptoms of Parkinson's disease occurred, a change in medication used to treat motor and/or non-motor symptoms of Parkinson's disease occurred and/or data was collected at a visit performed out of window when the participant was not treating when protocol requires (Present, Not Present).

#### 7.10.8. Other

Nonparametric tests that are not impacted by reasons for missing data will also be applied. In this case, only those that completed the study will be evaluated. If attrition in the active treatment arm significantly exceeds that of the passive treatment arm, treatment effects will be evaluated by comparing the active treatment study completers to the best responders of the passive treatment (of equal percentage). These sensitivity analyses will be used to give

greater confidence in the primary outcome and the combined measure of MDS-UPDRS Parts I, II, and III score.

## 7.11. ADDITIONAL SUPPORTING ANALYSES

Additional exploratory analyses that will be conducted to support clinical adoption are defined within the appendices to the Statistical Analysis Plan for OLE Study (ID: SNS-PD-003).

#### 8. REFERENCES

Administration\_CDRH, F. a. D. (2016). "Adaptive Designs for Medical Device Clinical Studies Guidance for Industry and Food and Drug Administration Staff."

Anderson, S. F., K. Kelley and S. E. Maxwell (2017). "Sample-Size Planning for More Accurate Statistical Power: A Method Adjusting Sample Effect Sizes for Publication Bias and Uncertainty." <a href="Psychol Sci 28(11)">Psychol Sci 28(11)</a>: 1547-1562.

Black, R., Rogers, L., Nicoletto, H., Adkins, H., Laskowitz, D. (2016). "Non-invasive neuromodulation using time-varying caloric vestibular stimulation - abstract." Headache **56**(S1).

Bloem, B. R., J. Marinus, Q. Almeida, L. Dibble, A. Nieuwboer, B. Post, E. Ruzicka, C. Goetz, G. Stebbins, P. Martinez-Martin, A. Schrag and C. Movement Disorders Society Rating Scales (2016). "Measurement instruments to assess posture, gait, and balance in Parkinson's disease: Critique and recommendations." <u>Mov Disord</u> **31**(9): 1342-1355.

Busner, J. and S. D. Targum (2007). "The clinical global impressions scale: applying a research tool in clinical practice." <u>Psychiatry (Edgmont)</u> **4**(7): 28-37.

Chaudhuri, K. R., A. Schrag, D. Weintraub, A. Rizos, C. Rodriguez-Blazquez, E. Mamikonyan and P. Martinez-Martin (2019). "The movement disorder society nonmotor rating scale: Initial validation study." <u>Mov Disord</u>.

Chaudhuri, K. R., Schrag, A., Weintraub, D., Rizos, A., Rodriguez-Basquez, C., Mamikonyan, E., Martinez-Martin, P. (2020). "The Movement Disorder Society Nonmotor Rating Scale: Initial Validation Study." <u>Movement Disorders</u> **35**(1): 17.

Christensen, M. C., M. Adair, H. Loft and R. S. McIntyre (2023). "The Motivation and Energy Inventory (MEI): Analysis of the clinically relevant response threshold in patients with major depressive disorder and emotional blunting using data from the COMPLETE study." J Affect Disord 323: 547-553.

Czobor, P., B. Sebe, K. Acsai, A. Barabassy, I. Laszlovszky, G. Nemeth, T. A. Furukawa and S. Leucht (2022). "What Is the Minimum Clinically Important Change in Negative Symptoms of Schizophrenia? PANSS Based Post-hoc Analyses of a Phase III Clinical Trial." <u>Front Psychiatry</u> 13: 816339.

Falissard, B., C. Sapin, J. Y. Loze, W. Landsberg and K. Hansen (2016). "Defining the minimal clinically important difference (MCID) of the Heinrichs-carpenter quality of life scale (QLS)." <u>Int J Methods Psychiatr Res</u> **25**(2): 101-111.

Ganju, J. and D. Rom (2017). "Non-inferiority versus superiority drug claims: the (not so) subtle distinction." <u>Trials</u> **18**(1): 278.

Godi, M., F. Franchignoni, M. Caligari, A. Giordano, A. M. Turcato and A. Nardone (2013). "Comparison of reliability, validity, and responsiveness of the mini-BESTest and Berg Balance Scale in patients with balance disorders." <u>Phys Ther</u> **93**(2): 158-167.

Goetz, C. G., S. Luo, L. Wang, B. C. Tilley, N. R. LaPelle and G. T. Stebbins (2015). "Handling missing values in the MDS-UPDRS." <u>Mov Disord</u> **30**(12): 1632-1638.

- Goetz, C. G., B. C. Tilley, S. R. Shaftman, G. T. Stebbins, S. Fahn, P. Martinez-Martin, W. Poewe, C. Sampaio, M. B. Stern, R. Dodel, B. Dubois, R. Holloway, J. Jankovic, J. Kulisevsky, A. E. Lang, A. Lees, S. Leurgans, P. A. LeWitt, D. Nyenhuis, C. W. Olanow, O. Rascol, A. Schrag, J. A. Teresi, J. J. van Hilten, N. LaPelle and U. R. T. F. Movement Disorder Society (2008). "Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS): scale presentation and clinimetric testing results." <u>Mov Disord</u> **23**(15): 2129-2170.
- Hauser, R. A., P. Auinger and G. Parkinson Study (2011). "Determination of minimal clinically important change in early and advanced Parkinson's disease." <u>Mov Disord</u> **26**(5): 813-818.
- Horvath, K., Z. Aschermann, P. Acs, G. Deli, J. Janszky, S. Komoly, E. Balazs, K. Takacs, K. Karadi and N. Kovacs (2015). "Minimal clinically important difference on the Motor Examination part of MDS-UPDRS." <u>Parkinsonism Relat Disord</u> **21**(12): 1421-1426.
- Horvath, K., Z. Aschermann, M. Kovacs, A. Makkos, M. Harmat, J. Janszky, S. Komoly, K. Karadi and N. Kovacs (2017). "Changes in Quality of Life in Parkinson's Disease: How Large Must They Be to Be Relevant?" <u>Neuroepidemiology</u> **48**(1-2): 1-8.
- Horvath, K., Z. Aschermann, M. Kovacs, A. Makkos, M. Harmat, J. Janszky, S. Komoly, K. Karadi and N. Kovacs (2017). "Minimal clinically important differences for the experiences of daily living parts of movement disorder society-sponsored unified Parkinson's disease rating scale." <u>Mov Disord</u> **32**(5): 789-793.
- Jenkinson, C., R. Fitzpatrick, V. Peto, R. Greenhall and N. Hyman (1997). "The Parkinson's Disease Questionnaire (PDQ-39): development and validation of a Parkinson's disease summary index score." Age Ageing 26(5): 353-357.
- Jost, S. T., M. A. Kaldenbach, A. Antonini, P. Martinez-Martin, L. Timmermann, P. Odin, R. Katzenschlager, R. Borgohain, A. Fasano, F. Stocchi, N. Hattori, P. L. Kukkle, M. Rodriguez-Violante, C. Falup-Pecurariu, S. Schade, J. N. Petry-Schmelzer, V. Metta, D. Weintraub, G. Deuschl, A. J. Espay, E. K. Tan, R. Bhidayasiri, V. S. C. Fung, F. Cardoso, C. Trenkwalder, P. Jenner, K. Ray Chaudhuri, H. S. Dafsari, P. International and G. Movement Disorders Society Non-Motor Parkinson Disease Study (2023). "Levodopa Dose Equivalency in Parkinson's Disease: Updated Systematic Review and Proposals." Mov Disord 38(7): 1236-1252.
- Kumar, R. and A. Indrayan (2011). "Receiver operating characteristic (ROC) curve for medical researchers." <u>Indian Pediatr</u> **48**(4): 277-287.
- Makkos, A., M. Kovacs, Z. Aschermann, M. Harmat, J. Janszky, K. Karadi and N. Kovacs (2018). "Are the MDS-UPDRS-Based Composite Scores Clinically Applicable?" <u>Mov Disord</u> **33**(5): 835-839.
- Norman, G. R., J. A. Sloan and K. W. Wyrwich (2003). "Interpretation of changes in health-related quality of life: the remarkable universality of half a standard deviation." <u>Med Care</u> **41**(5): 582-592.
- Rashid, W. G., M.K (2021). "A perspective of missing value imputation approaches." <u>Advances in Computational Intelligence and Communication Technology: Proceedings of CICT</u>: 307-315.
- Rubin, D. B., & Schenker, N. (1987). "Interval estimation from multiply-imputed data: a case study using census agriculture industry codes." <u>Journal of Official Statistics</u> **3**(4): 375.

Stebbins, G. T., C. G. Goetz, D. J. Burn, J. Jankovic, T. K. Khoo and B. C. Tilley (2013). "How to identify tremor dominant and postural instability/gait difficulty groups with the movement disorder society unified Parkinson's disease rating scale: comparison with the unified Parkinson's disease rating scale." <u>Mov Disord</u> **28**(5): 668-670.

van Wamelen, D. J., P. Martinez-Martin, D. Weintraub, A. Schrag, A. Antonini, C. Falup-Pecurariu, P. Odin, K. Ray Chaudhuri, P. International and G. Movement Disorder Society Parkinson's Disease Non-Motor Study (2021). "The Non-Motor Symptoms Scale in Parkinson's disease: Validation and use." <u>Acta Neurol Scand</u> **143**(1): 3-12.

Wilkinson, D., K. K. Ade, L. L. Rogers, D. K. Attix, M. Kuchibhatla, M. D. Slade, L. L. Smith, K. P. Poynter, D. T. Laskowitz, M. C. Freeman, M. E. Hoffer, J. R. Saper, D. L. Scott, M. Sakel, A. H. Calhoun and R. D. Black (2017). "Preventing Episodic Migraine With Caloric Vestibular Stimulation: A Randomized Controlled Trial." <u>Headache</u> 57(7): 1065-1087.

Wilkinson, D., A. Podlewska, S. E. Banducci, T. Pellat-Higgins, M. Slade, M. Bodani, M. Sakel, L. Smith, P. LeWitt and K. Ade (2019). "Caloric vestibular stimulation for the management of motor and non-motor symptoms in parkinson's disease: Intention-to-treat data." <u>Data Brief</u> 25: 104228.

Wilkinson, D., A. Podlewska, S. E. Banducci, T. Pellat-Higgins, M. Slade, M. Bodani, M. Sakel, L. Smith, P. LeWitt and K. K. Ade (2019). "Caloric vestibular stimulation for the management of motor and non-motor symptoms in Parkinson's disease." <u>Parkinsonism Relat Disord</u> **65**: 261-266.

Wilkinson, D., A. Podlewska and M. Sakel (2016). "A durable gain in motor and non-motor symptoms of Parkinson's Disease following repeated caloric vestibular stimulation: A single-case study." NeuroRehabilitation 38(2): 179-182.

Youden, W. J. (1950). "Index for rating diagnostic tests." Cancer 3(1): 32-35.

Yuan, Y. (2014). "Sensitivity analysis in multiple imputation for missing data." *Proceedings of the SAS Global Forum 2014 Conference*.

Zeger, S. L. and K. Y. Liang (1992). "An overview of methods for the analysis of longitudinal data." <u>Stat Med</u> **11**(14-15): 1825-1839.

Zorn, C. J. (2001). "Generalized estimating equation models for correlated data: A review with applications." <u>American Journal of Political Science</u> **45**(2).

# 9. APPENDICES

Appendix 1: STEM-PD RCT Schedule of Events

| | STEM-PD RCT | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessment | Screen<br>Study<br>Center | Baseline<br>1<br>Virtual | PC | PRO | Baseline 2 Study Center | PC | PRO | TX 1<br>Virtual | PC | PRO | TX 2<br>Virtual | PC | PRO | EOT<br>Study<br>Center |
| Day | -14 to -1 | 0<br>(+/- 3 days) | 15<br>(+/-<br>1<br>day) | 28<br>(+/- 1<br>day) | 29<br>(+/- 3 days | 43<br>(+/- 1<br>day) | 56<br>(+/- 1<br>day) | 57<br>(+/- 3<br>days) | 71<br>(+/- 1<br>day) | 84<br>(+/- 1<br>day) | 85<br>(+/- 3<br>days) | 99<br>(+/- 1<br>day) | 112<br>(+/- 1<br>day) | 113<br>(+/- 3 days) |
| Informed Consent | X | | | | | | | | | | | | | |
| Med Hx and ConMed<br>Hx Review | X | X | | | X | | | | | | | | | |
| Review<br>Inclusion/Exclusion | X | | | | X | | | | | | | | | |
| Pregnancy Test-Urine | | | | | X | | | | | | | | | |
| Educational Video and question/answer | | X | | | | | | | | | | | | |
| Ear Exam | X | | | | X | | | | | | | | | X |
| Height/Weight (height only at screen) | X | | | | X | | | | | | | | | X |
| MoCA | X | | | | X | | | | | | | | | X |

| | | | | | STEN | M-PD | RCT | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessment | Screen<br>Study<br>Center | Baseline<br>1<br>Virtual | PC | PRO | Baseline 2 Study Center | PC | PRO | TX1<br>Virtual | PC | PRO | TX2<br>Virtual | PC | PRO | EOT<br>Study<br>Center |
| Day | -14 to -1 | 0<br>(+/- 3 days) | 15<br>(+/- 1<br>day) | 28<br>(+/- 1<br>day) | 29<br>(+/- 3 days | 43<br>(+/- 1<br>day) | 56<br>(+/- 1<br>day) | 57 (+/- 3 days) | 71<br>(+/- 1<br>day) | 84<br>(+/- 1<br>day) | 85<br>(+/- 3<br>days) | 99<br>(+/- 1<br>day) | 112<br>(+/- 1 day) | 113<br>(+/- 3 days) |
| C-SSRS | X | | | | | | | | | | | | | |
| UPDRS I | | | | | X | | | | | | | | | X |
| MDS-UPDRS I | X | | | | X | | | | | | | | | X |
| MDS-NMS | | X | | | X NMF | | | X | | | X | | | X NMF |
| MDS-UPDRS II | | X | | X | | | X | | | X | | | X | |
| MDS-UPDRS III (onstate) | | X | | | X | | | X | | | X | | | X |
| Mini-BESTest | | | | | X | | | | | | | | | X |
| 10m TUG | | | | | X | | | | | | | | | X |
| 3m TUG & Finger<br>tapping (Encephalog<br>tests) | | | | | | | | X* | | | | | | |
| PDQ-39 | | X | | X | | | X | | | X | | | X | |
| Modified Schwab &<br>England | | | | | X | | | | | | | | | X |
| Pro-PD | X | | | | X | | | | | | | | | X |

| | | | | | STEN | M-PD | RCT | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessment | Screen<br>Study<br>Center | Baseline<br>1<br>Virtual | PC | PRO | Baseline 2 Study Center | PC | PRO | TX1<br>Virtual | PC | PRO | TX2<br>Virtual | PC | PRO | EOT<br>Study<br>Center |
| Day | -14 to -1 | 0<br>(+/- 3 days) | 15<br>(+/- 1<br>day) | 28<br>(+/- 1<br>day) | 29<br>(+/- 3 days | 43<br>(+/- 1<br>day) | 56<br>(+/- 1<br>day) | 57<br>(+/- 3 days) | 71<br>(+/- 1<br>day) | 84<br>(+/- 1<br>day) | 85<br>(+/- 3<br>days) | 99<br>(+/- 1<br>day) | 112<br>(+/- 1 day) | 113<br>(+/- 3 days) |
| oSDMT | | | | | X | | | | | | | | | X |
| PDSS-2 | | | | X | | | | | | | | | X | |
| ESS | | | | X | | | | | | | | | X | |
| PAS | | | | X | | | | | | | | | X | |
| FACIT-F | | | | X | | | | | | | | | X | |
| GDS | | | | X | | | | | | | | | X | |
| Transition<br>Questionnaire | | | | | | | X | | | | | | | |
| CGI-I (overall and focused) | | | | | X | | | | | | | | | X |
| UPDRS IV | | | | | X | | | | | | | | | X |
| Zarit Burden<br>Interview | | | | | X | | | | | | | | | X |
| Device Usability<br>Questionnaire | | | | | | | | | | | | | | X |
| Unpowered Device<br>Fitting | | | | | X | | | | | | | | | |

| | | | | | STEN | /I-PD | RCT | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessment | Screen<br>Study<br>Center | Baseline<br>1<br>Virtual | PC | PRO | Baseline 2 Study Center | PC | PRO | TX1<br>Virtual | PC | PRO | TX2<br>Virtual | PC | PRO | EOT<br>Study<br>Center |
| Day | -14 to -1 | 0<br>(+/- 3 days) | 15<br>(+/- 1<br>day) | 28<br>(+/- 1<br>day) | 29<br>(+/- 3 days | 43<br>(+/- 1<br>day) | 56<br>(+/- 1<br>day) | 57<br>(+/- 3 days) | 71<br>(+/- 1<br>day) | 84<br>(+/- 1<br>day) | 85<br>(+/- 3<br>days) | 99<br>(+/- 1<br>day) | 112<br>(+/- 1 day) | 113<br>(+/- 3 days) |
| Device Randomization and Training | | | | | X | | | | | | | | | |
| Device Return | | | | | | | | | | | | | | X |
| Home Assessment and ePRO Training | X | | | | | | | | | | | | | |
| Con Med & AE<br>Review | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Visit Scheduling and<br>Assessment Review | X | X | | | X | | | | | | | X | | |
| Treatment PeriodXX | | | | | | | | | | | | | | |
| X performed twice a day | X performed twice a day | | | | | | | | | | | | | |
| X* performed weekly | | | | | | | | | | | | | | |

# STEM-PD RCT SAP Appendix 2

This appendix provides instructions for creating the curves to interpret pooled interim analysis to evaluate the percent change in the coefficient of variation in the outcome that may be interpreted as the percent confidence that statistical significance of the outcome will be achieved in the study.

- 1. Determine baseline value of  $(SD / \overline{x})$ :  $(SD / \overline{x})_0$
- 2. Pick a percent increase in  $(SD / \overline{x})_0$
- 3. Calculate  $(SD/\overline{x})_1$ : Multiply  $(SD/\overline{x})_0$  by (1 + (percent increase / 100))

$$[(n-1)((SD/\bar{x})_0)^2]$$

4. Calculate  $\chi^2$ :  $\chi^2 = \frac{((SD/\overline{x})_1)^2}{((SD/\overline{x})_1)^2}$ 

- 5. Calculate right tailed probability, p, based on  $\chi^2$  and (n-1) degrees of freedom.
- 6. Calculate the measure of confidence: %Confidence = (1 p)

where:

SD = Standard Deviation

 $\overline{\mathbf{x}} = \mathbf{mean}$ 

n = number of subjects

p = right tailed probability

 $\chi$ 2 = Chi Square statistic

Subscript 0 denotes baseline

Subscript 1 denotes end of treatment

# **Interim Analysis Confidence Tables**

Alpha = 0.05

| n | 5% increas | e in stdev | $\chi^2$ | p | %<br>Confidence |
|---|---|---|---|---|---|
| | $(s/\overline{x})_0$ | $(s/\overline{x})_1$ | | | |
| 5 | 0.05 | 0.0525 | 3.6281 | 0.5413 | 45.8667 |
| 6 | 0.05 | 0.0525 | 4.5351 | 0.5248 | 47.5195 |
| 7 | 0.05 | 0.0525 | 5.4422 | 0.5115 | 48.8473 |
| 8 | 0.05 | 0.0525 | 6.3492 | 0.5004 | 49.9616 |
| 9 | 0.05 | 0.0525 | 7.2562 | 0.4907 | 50.9256 |
| 10 | 0.05 | 0.0525 | 8.1633 | 0.4822 | 51.7781 |
| 11 | 0.05 | 0.0525 | 9.0703 | 0.4746 | 52.5446 |
| 12 | 0.05 | 0.0525 | 9.9773 | 0.4676 | 53.2428 |
| 13 | 0.05 | 0.0525 | 10.8844 | 0.4611 | 53.8855 |
| 14 | 0.05 | 0.0525 | 11.7914 | 0.4552 | 54.4820 |
| 15 | 0.05 | 0.0525 | 12.6984 | 0.4496 | 55.0396 |
| 16 | 0.05 | 0.0525 | 13.6054 | 0.4444 | 55.5639 |
| 17 | 0.05 | 0.0525 | 14.5125 | 0.4394 | 56.0593 |
| 18 | 0.05 | 0.0525 | 15.4195 | 0.4347 | 56.5293 |
| 19 | 0.05 | 0.0525 | 16.3265 | 0.4302 | 56.9770 |
| 20 | 0.05 | 0.0525 | 17.2336 | 0.4260 | 57.4048 |
| 21 | 0.05 | 0.0525 | 18.1406 | 0.4219 | 57.8147 |
| 22 | 0.05 | 0.0525 | 19.0476 | 0.4179 | 58.2085 |

| 23 | 0.05 | 0.0525 | 19.9546 | 0.4141 | 58.5877 |
|----|------|--------|---------|--------|---------|
| 24 | 0.05 | 0.0525 | 20.8617 | 0.4105 | 58.9534 |
| 25 | 0.05 | 0.0525 | 21.7687 | 0.4069 | 59.3070 |
| 26 | 0.05 | 0.0525 | 22.6757 | 0.4035 | 59.6492 |
| 27 | 0.05 | 0.0525 | 23.5828 | 0.4002 | 59.9810 |
| 28 | 0.05 | 0.0525 | 24.4898 | 0.3970 | 60.3031 |
| 29 | 0.05 | 0.0525 | 25.3968 | 0.3938 | 60.6162 |
| 30 | 0.05 | 0.0525 | 26.3039 | 0.3908 | 60.9209 |
| 31 | 0.05 | 0.0525 | 27.2109 | 0.3878 | 61.2177 |
| 32 | 0.05 | 0.0525 | 28.1179 | 0.3849 | 61.5071 |
| 33 | 0.05 | 0.0525 | 29.0249 | 0.3821 | 61.7896 |
| 34 | 0.05 | 0.0525 | 29.9320 | 0.3793 | 62.0655 |
| 35 | 0.05 | 0.0525 | 30.8390 | 0.3766 | 62.3353 |
| 36 | 0.05 | 0.0525 | 31.7460 | 0.3740 | 62.5992 |
| 37 | 0.05 | 0.0525 | 32.6531 | 0.3714 | 62.8575 |
| 38 | 0.05 | 0.0525 | 33.5601 | 0.3689 | 63.1105 |
| 39 | 0.05 | 0.0525 | 34.4671 | 0.3664 | 63.3585 |
| 40 | 0.05 | 0.0525 | 35.3741 | 0.3640 | 63.6017 |
| 41 | 0.05 | 0.0525 | 36.2812 | 0.3616 | 63.8403 |
| 42 | 0.05 | 0.0525 | 37.1882 | 0.3593 | 64.0746 |
| 43 | 0.05 | 0.0525 | 38.0952 | 0.3570 | 64.3047 |
| 44 | 0.05 | 0.0525 | 39.0023 | 0.3547 | 64.5308 |
| 45 | 0.05 | 0.0525 | 39.9093 | 0.3525 | 64.7530 |

| 46 | 0.05 | 0.0525 | 40.8163 | 0.3503 | 64.9716 |
|----|------|--------|---------|--------|---------|
| 47 | 0.05 | 0.0525 | 41.7234 | 0.3481 | 65.1866 |
| 48 | 0.05 | 0.0525 | 42.6304 | 0.3460 | 65.3981 |
| 49 | 0.05 | 0.0525 | 43.5374 | 0.3439 | 65.6064 |
| 50 | 0.05 | 0.0525 | 44.4444 | 0.3419 | 65.8116 |
| 51 | 0.05 | 0.0525 | 45.3515 | 0.3399 | 66.0136 |
| 52 | 0.05 | 0.0525 | 46.2585 | 0.3379 | 66.2127 |
| 53 | 0.05 | 0.0525 | 47.1655 | 0.3359 | 66.4090 |
| 54 | 0.05 | 0.0525 | 48.0726 | 0.3340 | 66.6025 |
| 55 | 0.05 | 0.0525 | 48.9796 | 0.3321 | 66.7933 |
| 56 | 0.05 | 0.0525 | 49.8866 | 0.3302 | 66.9815 |
| 57 | 0.05 | 0.0525 | 50.7937 | 0.3283 | 67.1672 |
| 58 | 0.05 | 0.0525 | 51.7007 | 0.3265 | 67.3505 |
| 59 | 0.05 | 0.0525 | 52.6077 | 0.3247 | 67.5314 |
| 60 | 0.05 | 0.0525 | 53.5147 | 0.3229 | 67.7101 |
| 61 | 0.05 | 0.0525 | 54.4218 | 0.3211 | 67.8865 |
| 62 | 0.05 | 0.0525 | 55.3288 | 0.3194 | 68.0607 |
| 63 | 0.05 | 0.0525 | 56.2358 | 0.3177 | 68.2328 |
| 64 | 0.05 | 0.0525 | 57.1429 | 0.3160 | 68.4029 |
| 65 | 0.05 | 0.0525 | 58.0499 | 0.3143 | 68.5710 |
| 66 | 0.05 | 0.0525 | 58.9569 | 0.3126 | 68.7371 |
| 67 | 0.05 | 0.0525 | 59.8639 | 0.3110 | 68.9014 |
| 68 | 0.05 | 0.0525 | 60.7710 | 0.3094 | 69.0638 |

| 69 | 0.05 | 0.0525 | 61.6780 | 0.3078 | 69.2244 |
|----|------|--------|---------|--------|---------|
| 70 | 0.05 | 0.0525 | 62.5850 | 0.3062 | 69.3832 |
| 71 | 0.05 | 0.0525 | 63.4921 | 0.3046 | 69.5403 |
| 72 | 0.05 | 0.0525 | 64.3991 | 0.3030 | 69.6958 |
| 73 | 0.05 | 0.0525 | 65.3061 | 0.3015 | 69.8496 |
| 74 | 0.05 | 0.0525 | 66.2132 | 0.3000 | 70.0018 |
| 75 | 0.05 | 0.0525 | 67.1202 | 0.2985 | 70.1524 |

| | 10% increa | se in stdev | 2 | | % |
|---|---|---|---|---|---|
| n | $(s/\overline{x})_0$ | $(s/\overline{x})_1$ | $\chi^2$ | p | Confidence |
| 5 | 0.05 | 0.055 | 3.3058 | 0.4920 | 50.8016 |
| 6 | 0.05 | 0.055 | 4.1322 | 0.4695 | 53.0539 |
| 7 | 0.05 | 0.055 | 4.9587 | 0.4509 | 54.9124 |
| 8 | 0.05 | 0.055 | 5.7851 | 0.4349 | 56.5052 |
| 9 | 0.05 | 0.055 | 6.6116 | 0.4209 | 57.9061 |
| 10 | 0.05 | 0.055 | 7.4380 | 0.4084 | 59.1614 |
| 11 | 0.05 | 0.055 | 8.2645 | 0.3970 | 60.3022 |
| 12 | 0.05 | 0.055 | 9.0909 | 0.3865 | 61.3501 |
| 13 | 0.05 | 0.055 | 9.9174 | 0.3768 | 62.3211 |
| 14 | 0.05 | 0.055 | 10.7438 | 0.3677 | 63.2270 |
| 15 | 0.05 | 0.055 | 11.5702 | 0.3592 | 64.0772 |
| 16 | 0.05 | 0.055 | 12.3967 | 0.3512 | 64.8788 |
| 17 | 0.05 | 0.055 | 13.2231 | 0.3436 | 65.6378 |
| 18 | 0.05 | 0.055 | 14.0496 | 0.3364 | 66.3589 |
| 19 | 0.05 | 0.055 | 14.8760 | 0.3295 | 67.0461 |
| 20 | 0.05 | 0.055 | 15.7025 | 0.3230 | 67.7027 |
| 21 | 0.05 | 0.055 | 16.5289 | 0.3167 | 68.3316 |
| 22 | 0.05 | 0.055 | 17.3554 | 0.3106 | 68.9352 |
| 23 | 0.05 | 0.055 | 18.1818 | 0.3048 | 69.5156 |
| 24 | 0.05 | 0.055 | 19.0083 | 0.2993 | 70.0745 |

| 25 | 0.05 | 0.055 | 19.8347 | 0.2939 | 70.6136 |
|----|------|-------|---------|--------|---------|
| 26 | 0.05 | 0.055 | 20.6612 | 0.2887 | 71.1343 |
| 27 | 0.05 | 0.055 | 21.4876 | 0.2836 | 71.6378 |
| 28 | 0.05 | 0.055 | 22.3140 | 0.2787 | 72.1253 |
| 29 | 0.05 | 0.055 | 23.1405 | 0.2740 | 72.5977 |
| 30 | 0.05 | 0.055 | 23.9669 | 0.2694 | 73.0560 |
| 31 | 0.05 | 0.055 | 24.7934 | 0.2650 | 73.5009 |
| 32 | 0.05 | 0.055 | 25.6198 | 0.2607 | 73.9333 |
| 33 | 0.05 | 0.055 | 26.4463 | 0.2565 | 74.3536 |
| 34 | 0.05 | 0.055 | 27.2727 | 0.2524 | 74.7627 |
| 35 | 0.05 | 0.055 | 28.0992 | 0.2484 | 75.1611 |
| 36 | 0.05 | 0.055 | 28.9256 | 0.2445 | 75.5491 |
| 37 | 0.05 | 0.055 | 29.7521 | 0.2407 | 75.9275 |
| 38 | 0.05 | 0.055 | 30.5785 | 0.2370 | 76.2965 |
| 39 | 0.05 | 0.055 | 31.4050 | 0.2334 | 76.6566 |
| 40 | 0.05 | 0.055 | 32.2314 | 0.2299 | 77.0082 |
| 41 | 0.05 | 0.055 | 33.0579 | 0.2265 | 77.3517 |
| 42 | 0.05 | 0.055 | 33.8843 | 0.2231 | 77.6873 |
| 43 | 0.05 | 0.055 | 34.7107 | 0.2198 | 78.0154 |
| 44 | 0.05 | 0.055 | 35.5372 | 0.2166 | 78.3362 |
| 45 | 0.05 | 0.055 | 36.3636 | 0.2135 | 78.6501 |
| 46 | 0.05 | 0.055 | 37.1901 | 0.2104 | 78.9573 |
| 47 | 0.05 | 0.055 | 38.0165 | 0.2074 | 79.2580 |

| 48 | 0.05 | 0.055 | 38.8430 | 0.2045 | 79.5524 |
|----|------|-------|---------|--------|---------|
| 49 | 0.05 | 0.055 | 39.6694 | 0.2016 | 79.8409 |
| 50 | 0.05 | 0.055 | 40.4959 | 0.1988 | 80.1235 |
| 51 | 0.05 | 0.055 | 41.3223 | 0.1960 | 80.4005 |
| 52 | 0.05 | 0.055 | 42.1488 | 0.1933 | 80.6721 |
| 53 | 0.05 | 0.055 | 42.9752 | 0.1906 | 80.9383 |
| 54 | 0.05 | 0.055 | 43.8017 | 0.1880 | 81.1995 |
| 55 | 0.05 | 0.055 | 44.6281 | 0.1854 | 81.4557 |
| 56 | 0.05 | 0.055 | 45.4545 | 0.1829 | 81.7071 |
| 57 | 0.05 | 0.055 | 46.2810 | 0.1805 | 81.9539 |
| 58 | 0.05 | 0.055 | 47.1074 | 0.1780 | 82.1961 |
| 59 | 0.05 | 0.055 | 47.9339 | 0.1757 | 82.4339 |
| 60 | 0.05 | 0.055 | 48.7603 | 0.1733 | 82.6674 |
| 61 | 0.05 | 0.055 | 49.5868 | 0.1710 | 82.8968 |
| 62 | 0.05 | 0.055 | 50.4132 | 0.1688 | 83.1221 |
| 63 | 0.05 | 0.055 | 51.2397 | 0.1666 | 83.3435 |
| 64 | 0.05 | 0.055 | 52.0661 | 0.1644 | 83.5610 |
| 65 | 0.05 | 0.055 | 52.8926 | 0.1623 | 83.7749 |
| 66 | 0.05 | 0.055 | 53.7190 | 0.1601 | 83.9850 |
| 67 | 0.05 | 0.055 | 54.5455 | 0.1581 | 84.1917 |
| 68 | 0.05 | 0.055 | 55.3719 | 0.1561 | 84.3948 |
| 69 | 0.05 | 0.055 | 56.1983 | 0.1541 | 84.5946 |
| 70 | 0.05 | 0.055 | 57.0248 | 0.1521 | 84.7911 |
| 71 | 0.05 | 0.055 | 57.8512 | 0.1502 | 84.9844 |
|----|------|-------|---------|--------|---------|
| 72 | 0.05 | 0.055 | 58.6777 | 0.1483 | 85.1746 |
| 73 | 0.05 | 0.055 | 59.5041 | 0.1464 | 85.3617 |
| 74 | 0.05 | 0.055 | 60.3306 | 0.1445 | 85.5458 |
| 75 | 0.05 | 0.055 | 61.1570 | 0.1427 | 85.7269 |

| n | 15% increa | se in stdev | $\chi^2$ | n | % |
|---|---|---|---|---|---|
| n | $(s/\overline{x})_0$ | $(s/\overline{x})_1$ | χ | p | Confidence |
| 5 | 0.05 | 0.0575 | 3.0246 | 0.4463 | 55.3721 |
| 6 | 0.05 | 0.0575 | 3.7807 | 0.4186 | 58.1399 |
| 7 | 0.05 | 0.0575 | 4.5369 | 0.3956 | 60.4427 |
| 8 | 0.05 | 0.0575 | 5.2930 | 0.3757 | 62.4254 |
| 9 | 0.05 | 0.0575 | 6.0491 | 0.3583 | 64.1726 |
| 10 | 0.05 | 0.0575 | 6.8053 | 0.3426 | 65.7383 |
| 11 | 0.05 | 0.0575 | 7.5614 | 0.3284 | 67.1589 |
| 12 | 0.05 | 0.0575 | 8.3176 | 0.3154 | 68.4605 |
| 13 | 0.05 | 0.0575 | 9.0737 | 0.3034 | 69.6621 |
| 14 | 0.05 | 0.0575 | 9.8299 | 0.2922 | 70.7784 |
| 15 | 0.05 | 0.0575 | 10.5860 | 0.2818 | 71.8208 |
| 16 | 0.05 | 0.0575 | 11.3422 | 0.2720 | 72.7984 |
| 17 | 0.05 | 0.0575 | 12.0983 | 0.2628 | 73.7186 |
| 18 | 0.05 | 0.0575 | 12.8544 | 0.2541 | 74.5874 |
| 19 | 0.05 | 0.0575 | 13.6106 | 0.2459 | 75.4101 |
| 20 | 0.05 | 0.0575 | 14.3667 | 0.2381 | 76.1908 |
| 21 | 0.05 | 0.0575 | 15.1229 | 0.2307 | 76.9334 |
| 22 | 0.05 | 0.0575 | 15.8790 | 0.2236 | 77.6410 |
| 23 | 0.05 | 0.0575 | 16.6352 | 0.2168 | 78.3163 |
| 24 | 0.05 | 0.0575 | 17.3913 | 0.2104 | 78.9619 |

| 25 | 0.05 | 0.0575 | 18.1474 | 0.2042 | 79.5798 |
|----|------|--------|---------|--------|---------|
| 26 | 0.05 | 0.0575 | 18.9036 | 0.1983 | 80.1720 |
| 27 | 0.05 | 0.0575 | 19.6597 | 0.1926 | 80.7401 |
| 28 | 0.05 | 0.0575 | 20.4159 | 0.1871 | 81.2858 |
| 29 | 0.05 | 0.0575 | 21.1720 | 0.1819 | 81.8104 |
| 30 | 0.05 | 0.0575 | 21.9282 | 0.1768 | 82.3152 |
| 31 | 0.05 | 0.0575 | 22.6843 | 0.1720 | 82.8012 |
| 32 | 0.05 | 0.0575 | 23.4405 | 0.1673 | 83.2696 |
| 33 | 0.05 | 0.0575 | 24.1966 | 0.1628 | 83.7213 |
| 34 | 0.05 | 0.0575 | 24.9527 | 0.1584 | 84.1571 |
| 35 | 0.05 | 0.0575 | 25.7089 | 0.1542 | 84.5780 |
| 36 | 0.05 | 0.0575 | 26.4650 | 0.1502 | 84.9845 |
| 37 | 0.05 | 0.0575 | 27.2212 | 0.1462 | 85.3775 |
| 38 | 0.05 | 0.0575 | 27.9773 | 0.1424 | 85.7575 |
| 39 | 0.05 | 0.0575 | 28.7335 | 0.1387 | 86.1252 |
| 40 | 0.05 | 0.0575 | 29.4896 | 0.1352 | 86.4811 |
| 41 | 0.05 | 0.0575 | 30.2457 | 0.1317 | 86.8257 |
| 42 | 0.05 | 0.0575 | 31.0019 | 0.1284 | 87.1595 |
| 43 | 0.05 | 0.0575 | 31.7580 | 0.1252 | 87.4831 |
| 44 | 0.05 | 0.0575 | 32.5142 | 0.1220 | 87.7967 |
| 45 | 0.05 | 0.0575 | 33.2703 | 0.1190 | 88.1009 |
| 46 | 0.05 | 0.0575 | 34.0265 | 0.1160 | 88.3959 |
| 47 | 0.05 | 0.0575 | 34.7826 | 0.1132 | 88.6822 |

| 48 | 0.05 | 0.0575 | 35.5388 | 0.1104 | 88.9601 |
|----|------|--------|---------|--------|---------|
| 49 | 0.05 | 0.0575 | 36.2949 | 0.1077 | 89.2299 |
| 50 | 0.05 | 0.0575 | 37.0510 | 0.1051 | 89.4920 |
| 51 | 0.05 | 0.0575 | 37.8072 | 0.1025 | 89.7465 |
| 52 | 0.05 | 0.0575 | 38.5633 | 0.1001 | 89.9938 |
| 53 | 0.05 | 0.0575 | 39.3195 | 0.0977 | 90.2342 |
| 54 | 0.05 | 0.0575 | 40.0756 | 0.0953 | 90.4679 |
| 55 | 0.05 | 0.0575 | 40.8318 | 0.0930 | 90.6950 |
| 56 | 0.05 | 0.0575 | 41.5879 | 0.0908 | 90.9160 |
| 57 | 0.05 | 0.0575 | 42.3440 | 0.0887 | 91.1309 |
| 58 | 0.05 | 0.0575 | 43.1002 | 0.0866 | 91.3399 |
| 59 | 0.05 | 0.0575 | 43.8563 | 0.0846 | 91.5434 |
| 60 | 0.05 | 0.0575 | 44.6125 | 0.0826 | 91.7413 |
| 61 | 0.05 | 0.0575 | 45.3686 | 0.0807 | 91.9340 |
| 62 | 0.05 | 0.0575 | 46.1248 | 0.0788 | 92.1217 |
| 63 | 0.05 | 0.0575 | 46.8809 | 0.0770 | 92.3043 |
| 64 | 0.05 | 0.0575 | 47.6371 | 0.0752 | 92.4822 |
| 65 | 0.05 | 0.0575 | 48.3932 | 0.0734 | 92.6555 |
| 66 | 0.05 | 0.0575 | 49.1493 | 0.0718 | 92.8243 |
| 67 | 0.05 | 0.0575 | 49.9055 | 0.0701 | 92.9887 |
| 68 | 0.05 | 0.0575 | 50.6616 | 0.0685 | 93.1489 |
| 69 | 0.05 | 0.0575 | 51.4178 | 0.0669 | 93.3051 |
| 70 | 0.05 | 0.0575 | 52.1739 | 0.0654 | 93.4573 |

| 71 | 0.05 | 0.0575 | 52.9301 | 0.0639 | 93.6056 |
|----|------|--------|---------|--------|---------|
| 72 | 0.05 | 0.0575 | 53.6862 | 0.0625 | 93.7502 |
| 73 | 0.05 | 0.0575 | 54.4423 | 0.0611 | 93.8912 |
| 74 | 0.05 | 0.0575 | 55.1985 | 0.0597 | 94.0287 |
| 75 | 0.05 | 0.0575 | 55.9546 | 0.0584 | 94.1627 |

| n | 20% increa | ase in stdev | $\chi^2$ | n | % |
|---|---|---|---|---|---|
| n | $(s/\overline{x})_0$ | $(s/\overline{x})_1$ | χ | p | Confidence |
| 5 | 0.05 | 0.06 | 2.7778 | 0.4043 | 59.5675 |
| 6 | 0.05 | 0.06 | 3.4722 | 0.3724 | 62.7595 |
| 7 | 0.05 | 0.06 | 4.1667 | 0.3459 | 65.4133 |
| 8 | 0.05 | 0.06 | 4.8611 | 0.3231 | 67.6908 |
| 9 | 0.05 | 0.06 | 5.5556 | 0.3031 | 69.6877 |
| 10 | 0.05 | 0.06 | 6.2500 | 0.2853 | 71.4660 |
| 11 | 0.05 | 0.06 | 6.9444 | 0.2693 | 73.0679 |
| 12 | 0.05 | 0.06 | 7.6389 | 0.2548 | 74.5240 |
| 13 | 0.05 | 0.06 | 8.3333 | 0.2414 | 75.8569 |
| 14 | 0.05 | 0.06 | 9.0278 | 0.2292 | 77.0842 |
| 15 | 0.05 | 0.06 | 9.7222 | 0.2178 | 78.2197 |
| 16 | 0.05 | 0.06 | 10.4167 | 0.2073 | 79.2745 |
| 17 | 0.05 | 0.06 | 11.1111 | 0.1974 | 80.2576 |
| 18 | 0.05 | 0.06 | 11.8056 | 0.1882 | 81.1766 |
| 19 | 0.05 | 0.06 | 12.5000 | 0.1796 | 82.0379 |
| 20 | 0.05 | 0.06 | 13.1944 | 0.1715 | 82.8470 |
| 21 | 0.05 | 0.06 | 13.8889 | 0.1639 | 83.6085 |
| 22 | 0.05 | 0.06 | 14.5833 | 0.1567 | 84.3264 |
| 23 | 0.05 | 0.06 | 15.2778 | 0.1500 | 85.0044 |
| 24 | 0.05 | 0.06 | 15.9722 | 0.1435 | 85.6455 |

| 25 | 0.05 | 0.06 | 16.6667 | 0.1375 | 86.2526 |
|----|------|------|---------|--------|---------|
| 26 | 0.05 | 0.06 | 17.3611 | 0.1317 | 86.8281 |
| 27 | 0.05 | 0.06 | 18.0556 | 0.1263 | 87.3743 |
| 28 | 0.05 | 0.06 | 18.7500 | 0.1211 | 87.8931 |
| 29 | 0.05 | 0.06 | 19.4444 | 0.1161 | 88.3864 |
| 30 | 0.05 | 0.06 | 20.1389 | 0.1114 | 88.8557 |
| 31 | 0.05 | 0.06 | 20.8333 | 0.1070 | 89.3027 |
| 32 | 0.05 | 0.06 | 21.5278 | 0.1027 | 89.7286 |
| 33 | 0.05 | 0.06 | 22.2222 | 0.0987 | 90.1348 |
| 34 | 0.05 | 0.06 | 22.9167 | 0.0948 | 90.5224 |
| 35 | 0.05 | 0.06 | 23.6111 | 0.0911 | 90.8924 |
| 36 | 0.05 | 0.06 | 24.3056 | 0.0875 | 91.2459 |
| 37 | 0.05 | 0.06 | 25.0000 | 0.0842 | 91.5837 |
| 38 | 0.05 | 0.06 | 25.6944 | 0.0809 | 91.9067 |
| 39 | 0.05 | 0.06 | 26.3889 | 0.0778 | 92.2156 |
| 40 | 0.05 | 0.06 | 27.0833 | 0.0749 | 92.5113 |
| 41 | 0.05 | 0.06 | 27.7778 | 0.0721 | 92.7944 |
| 42 | 0.05 | 0.06 | 28.4722 | 0.0693 | 93.0656 |
| 43 | 0.05 | 0.06 | 29.1667 | 0.0667 | 93.3254 |
| 44 | 0.05 | 0.06 | 29.8611 | 0.0643 | 93.5743 |
| 45 | 0.05 | 0.06 | 30.5556 | 0.0619 | 93.8130 |
| 46 | 0.05 | 0.06 | 31.2500 | 0.0596 | 94.0419 |
| 47 | 0.05 | 0.06 | 31.9444 | 0.0574 | 94.2615 |

| 48 | 0.05 | 0.06 | 32.6389 | 0.0553 | 94.4723 |
|----|------|------|---------|--------|---------|
| 49 | 0.05 | 0.06 | 33.3333 | 0.0533 | 94.6745 |
| 50 | 0.05 | 0.06 | 34.0278 | 0.0513 | 94.8687 |
| 51 | 0.05 | 0.06 | 34.7222 | 0.0494 | 95.0552 |
| 52 | 0.05 | 0.06 | 35.4167 | 0.0477 | 95.2343 |
| 53 | 0.05 | 0.06 | 36.1111 | 0.0459 | 95.4063 |
| 54 | 0.05 | 0.06 | 36.8056 | 0.0443 | 95.5717 |
| 55 | 0.05 | 0.06 | 37.5000 | 0.0427 | 95.7306 |
| 56 | 0.05 | 0.06 | 38.1944 | 0.0412 | 95.8834 |
| 57 | 0.05 | 0.06 | 38.8889 | 0.0397 | 96.0303 |
| 58 | 0.05 | 0.06 | 39.5833 | 0.0383 | 96.1716 |
| 59 | 0.05 | 0.06 | 40.2778 | 0.0369 | 96.3075 |
| 60 | 0.05 | 0.06 | 40.9722 | 0.0356 | 96.4383 |
| 61 | 0.05 | 0.06 | 41.6667 | 0.0344 | 96.5641 |
| 62 | 0.05 | 0.06 | 42.3611 | 0.0331 | 96.6851 |
| 63 | 0.05 | 0.06 | 43.0556 | 0.0320 | 96.8016 |
| 64 | 0.05 | 0.06 | 43.7500 | 0.0309 | 96.9138 |
| 65 | 0.05 | 0.06 | 44.4444 | 0.0298 | 97.0218 |
| 66 | 0.05 | 0.06 | 45.1389 | 0.0287 | 97.1258 |
| 67 | 0.05 | 0.06 | 45.8333 | 0.0277 | 97.2259 |
| 68 | 0.05 | 0.06 | 46.5278 | 0.0268 | 97.3224 |
| 69 | 0.05 | 0.06 | 47.2222 | 0.0258 | 97.4153 |
| 70 | 0.05 | 0.06 | 47.9167 | 0.0250 | 97.5048 |

| 71 | 0.05 | 0.06 | 48.6111 | 0.0241 | 97.5910 |
|----|------|------|---------|--------|---------|
| 72 | 0.05 | 0.06 | 49.3056 | 0.0233 | 97.6741 |
| 73 | 0.05 | 0.06 | 50.0000 | 0.0225 | 97.7542 |
| 74 | 0.05 | 0.06 | 50.6944 | 0.0217 | 97.8314 |
| 75 | 0.05 | 0.06 | 51.3889 | 0.0209 | 97.9058 |

| | 25% increa | se in stdev | 3.2000 0.3308 3.8400 0.3017 4.4800 0.2769 5.1200 0.2553 5.7600 0.2363 6.4000 0.2194 7.0400 0.2042 7.6800 0.1904 8.3200 0.1779 8.9600 0.1664 | - | % |
|---|---|---|---|---|---|
| n | $(s/\overline{x})_0$ | $(s/\overline{x})_1$ | χ- | þ | Confidence |
| 5 | 0.05 | 0.0625 | 2.5600 | 0.3661 | 63.3925 |
| 6 | 0.05 | 0.0625 | 3.2000 | 0.3308 | 66.9183 |
| 7 | 0.05 | 0.0625 | 3.8400 | 0.3017 | 69.8318 |
| 8 | 0.05 | 0.0625 | 4.4800 | 0.2769 | 72.3124 |
| 9 | 0.05 | 0.0625 | 5.1200 | 0.2553 | 74.4677 |
| 10 | 0.05 | 0.0625 | 5.7600 | 0.2363 | 76.3677 |
| 11 | 0.05 | 0.0625 | 6.4000 | 0.2194 | 78.0613 |
| 12 | 0.05 | 0.0625 | 7.0400 | 0.2042 | 79.5835 |
| 13 | 0.05 | 0.0625 | 7.6800 | 0.1904 | 80.9611 |
| 14 | 0.05 | 0.0625 | 8.3200 | 0.1779 | 82.2146 |
| 15 | 0.05 | 0.0625 | 8.9600 | 0.1664 | 83.3604 |
| 16 | 0.05 | 0.0625 | 9.6000 | 0.1559 | 84.4119 |
| 17 | 0.05 | 0.0625 | 10.2400 | 0.1462 | 85.3798 |
| 18 | 0.05 | 0.0625 | 10.8800 | 0.1373 | 86.2734 |
| 19 | 0.05 | 0.0625 | 11.5200 | 0.1290 | 87.1003 |
| 20 | 0.05 | 0.0625 | 12.1600 | 0.1213 | 87.8673 |
| 21 | 0.05 | 0.0625 | 12.8000 | 0.1142 | 88.5799 |
| 22 | 0.05 | 0.0625 | 13.4400 | 0.1076 | 89.2432 |
| 23 | 0.05 | 0.0625 | 14.0800 | 0.1014 | 89.8616 |
| 24 | 0.05 | 0.0625 | 14.7200 | 0.0956 | 90.4387 |

| 25 | 0.05 | 0.0625 | 15.3600 | 0.0902 | 90.9782 |
|----|------|--------|---------|--------|---------|
| 26 | 0.05 | 0.0625 | 16.0000 | 0.0852 | 91.4829 |
| 27 | 0.05 | 0.0625 | 16.6400 | 0.0804 | 91.9556 |
| 28 | 0.05 | 0.0625 | 17.2800 | 0.0760 | 92.3988 |
| 29 | 0.05 | 0.0625 | 17.9200 | 0.0719 | 92.8146 |
| 30 | 0.05 | 0.0625 | 18.5600 | 0.0679 | 93.2051 |
| 31 | 0.05 | 0.0625 | 19.2000 | 0.0643 | 93.5721 |
| 32 | 0.05 | 0.0625 | 19.8400 | 0.0608 | 93.9172 |
| 33 | 0.05 | 0.0625 | 20.4800 | 0.0576 | 94.2420 |
| 34 | 0.05 | 0.0625 | 21.1200 | 0.0545 | 94.5477 |
| 35 | 0.05 | 0.0625 | 21.7600 | 0.0516 | 94.8358 |
| 36 | 0.05 | 0.0625 | 22.4000 | 0.0489 | 95.1073 |
| 37 | 0.05 | 0.0625 | 23.0400 | 0.0464 | 95.3634 |
| 38 | 0.05 | 0.0625 | 23.6800 | 0.0440 | 95.6050 |
| 39 | 0.05 | 0.0625 | 24.3200 | 0.0417 | 95.8330 |
| 40 | 0.05 | 0.0625 | 24.9600 | 0.0395 | 96.0483 |
| 41 | 0.05 | 0.0625 | 25.6000 | 0.0375 | 96.2517 |
| 42 | 0.05 | 0.0625 | 26.2400 | 0.0356 | 96.4439 |
| 43 | 0.05 | 0.0625 | 26.8800 | 0.0337 | 96.6256 |
| 44 | 0.05 | 0.0625 | 27.5200 | 0.0320 | 96.7975 |
| 45 | 0.05 | 0.0625 | 28.1600 | 0.0304 | 96.9600 |
| 46 | 0.05 | 0.0625 | 28.8000 | 0.0289 | 97.1138 |
| 47 | 0.05 | 0.0625 | 29.4400 | 0.0274 | 97.2594 |

| 48 | 0.05 | 0.0625 | 30.0800 | 0.0260 | 97.3972 |
|----|------|--------|---------|--------|---------|
| 49 | 0.05 | 0.0625 | 30.7200 | 0.0247 | 97.5277 |
| 50 | 0.05 | 0.0625 | 31.3600 | 0.0235 | 97.6513 |
| 51 | 0.05 | 0.0625 | 32.0000 | 0.0223 | 97.7685 |
| 52 | 0.05 | 0.0625 | 32.6400 | 0.0212 | 97.8795 |
| 53 | 0.05 | 0.0625 | 33.2800 | 0.0202 | 97.9847 |
| 54 | 0.05 | 0.0625 | 33.9200 | 0.0192 | 98.0844 |
| 55 | 0.05 | 0.0625 | 34.5600 | 0.0182 | 98.1790 |
| 56 | 0.05 | 0.0625 | 35.2000 | 0.0173 | 98.2687 |
| 57 | 0.05 | 0.0625 | 35.8400 | 0.0165 | 98.3538 |
| 58 | 0.05 | 0.0625 | 36.4800 | 0.0157 | 98.4346 |
| 59 | 0.05 | 0.0625 | 37.1200 | 0.0149 | 98.5112 |
| 60 | 0.05 | 0.0625 | 37.7600 | 0.0142 | 98.5839 |
| 61 | 0.05 | 0.0625 | 38.4000 | 0.0135 | 98.6530 |
| 62 | 0.05 | 0.0625 | 39.0400 | 0.0128 | 98.7185 |
| 63 | 0.05 | 0.0625 | 39.6800 | 0.0122 | 98.7808 |
| 64 | 0.05 | 0.0625 | 40.3200 | 0.0116 | 98.8399 |
| 65 | 0.05 | 0.0625 | 40.9600 | 0.0110 | 98.8961 |
| 66 | 0.05 | 0.0625 | 41.6000 | 0.0105 | 98.9494 |
| 67 | 0.05 | 0.0625 | 42.2400 | 0.0100 | 99.0001 |
| 68 | 0.05 | 0.0625 | 42.8800 | 0.0095 | 99.0482 |
| 69 | 0.05 | 0.0625 | 43.5200 | 0.0091 | 99.0940 |
| 70 | 0.05 | 0.0625 | 44.1600 | 0.0086 | 99.1375 |

| 71 | 0.05 | 0.0625 | 44.8000 | 0.0082 | 99.1788 |
|----|------|--------|---------|--------|---------|
| 72 | 0.05 | 0.0625 | 45.4400 | 0.0078 | 99.2181 |
| 73 | 0.05 | 0.0625 | 46.0800 | 0.0074 | 99.2555 |
| 74 | 0.05 | 0.0625 | 46.7200 | 0.0071 | 99.2910 |
| 75 | 0.05 | 0.0625 | 47.3600 | 0.0068 | 99.3248 |

| n | 30% increa | 30% increase in stdev | | n | % |
|---|---|---|---|---|---|
| | $(s/\overline{x})_0$ | $(s/\overline{x})_1$ | $\chi^2$ | p | Confidence |
| 5 | 0.05 | 0.065 | 2.3669 | 0.3314 | 66.8624 |
| 6 | 0.05 | 0.065 | 2.9586 | 0.2936 | 70.6372 |
| 7 | 0.05 | 0.065 | 3.5503 | 0.2627 | 73.7266 |
| 8 | 0.05 | 0.065 | 4.1420 | 0.2367 | 76.3283 |
| 9 | 0.05 | 0.065 | 4.7337 | 0.2144 | 78.5620 |
| 10 | 0.05 | 0.065 | 5.3254 | 0.1949 | 80.5066 |
| 11 | 0.05 | 0.065 | 5.9172 | 0.1778 | 82.2174 |
| 12 | 0.05 | 0.065 | 6.5089 | 0.1627 | 83.7349 |
| 13 | 0.05 | 0.065 | 7.1006 | 0.1491 | 85.0895 |
| 14 | 0.05 | 0.065 | 7.6923 | 0.1369 | 86.3052 |
| 15 | 0.05 | 0.065 | 8.2840 | 0.1260 | 87.4010 |
| 16 | 0.05 | 0.065 | 8.8757 | 0.1161 | 88.3924 |
| 17 | 0.05 | 0.065 | 9.4675 | 0.1071 | 89.2922 |
| 18 | 0.05 | 0.065 | 10.0592 | 0.0989 | 90.1111 |
| 19 | 0.05 | 0.065 | 10.6509 | 0.0914 | 90.8580 |
| 20 | 0.05 | 0.065 | 11.2426 | 0.0846 | 91.5408 |
| 21 | 0.05 | 0.065 | 11.8343 | 0.0783 | 92.1661 |
| 22 | 0.05 | 0.065 | 12.4260 | 0.0726 | 92.7396 |
| 23 | 0.05 | 0.065 | 13.0178 | 0.0673 | 93.2665 |
| 24 | 0.05 | 0.065 | 13.6095 | 0.0625 | 93.7512 |

| 25 | 0.05 | 0.065 | 14.2012 | 0.0580 | 94.1975 |
|----|------|-------|---------|--------|---------|
| 26 | 0.05 | 0.065 | 14.7929 | 0.0539 | 94.6090 |
| 27 | 0.05 | 0.065 | 15.3846 | 0.0501 | 94.9888 |
| 28 | 0.05 | 0.065 | 15.9763 | 0.0466 | 95.3397 |
| 29 | 0.05 | 0.065 | 16.5680 | 0.0434 | 95.6640 |
| 30 | 0.05 | 0.065 | 17.1598 | 0.0404 | 95.9642 |
| 31 | 0.05 | 0.065 | 17.7515 | 0.0376 | 96.2420 |
| 32 | 0.05 | 0.065 | 18.3432 | 0.0350 | 96.4995 |
| 33 | 0.05 | 0.065 | 18.9349 | 0.0326 | 96.7382 |
| 34 | 0.05 | 0.065 | 19.5266 | 0.0304 | 96.9596 |
| 35 | 0.05 | 0.065 | 20.1183 | 0.0283 | 97.1651 |
| 36 | 0.05 | 0.065 | 20.7101 | 0.0264 | 97.3560 |
| 37 | 0.05 | 0.065 | 21.3018 | 0.0247 | 97.5333 |
| 38 | 0.05 | 0.065 | 21.8935 | 0.0230 | 97.6982 |
| 39 | 0.05 | 0.065 | 22.4852 | 0.0215 | 97.8514 |
| 40 | 0.05 | 0.065 | 23.0769 | 0.0201 | 97.9940 |
| 41 | 0.05 | 0.065 | 23.6686 | 0.0187 | 98.1267 |
| 42 | 0.05 | 0.065 | 24.2604 | 0.0175 | 98.2502 |
| 43 | 0.05 | 0.065 | 24.8521 | 0.0163 | 98.3653 |
| 44 | 0.05 | 0.065 | 25.4438 | 0.0153 | 98.4725 |
| 45 | 0.05 | 0.065 | 26.0355 | 0.0143 | 98.5724 |
| 46 | 0.05 | 0.065 | 26.6272 | 0.0133 | 98.6655 |
| 47 | 0.05 | 0.065 | 27.2189 | 0.0125 | 98.7523 |

| 48 | 0.05 | 0.065 | 27.8107 | 0.0117 | 98.8332 |
|----|------|-------|---------|--------|---------|
| 49 | 0.05 | 0.065 | 28.4024 | 0.0109 | 98.9088 |
| 50 | 0.05 | 0.065 | 28.9941 | 0.0102 | 98.9793 |
| 51 | 0.05 | 0.065 | 29.5858 | 0.0095 | 99.0450 |
| 52 | 0.05 | 0.065 | 30.1775 | 0.0089 | 99.1065 |
| 53 | 0.05 | 0.065 | 30.7692 | 0.0084 | 99.1638 |
| 54 | 0.05 | 0.065 | 31.3609 | 0.0078 | 99.2174 |
| 55 | 0.05 | 0.065 | 31.9527 | 0.0073 | 99.2674 |
| 56 | 0.05 | 0.065 | 32.5444 | 0.0069 | 99.3142 |
| 57 | 0.05 | 0.065 | 33.1361 | 0.0064 | 99.3578 |
| 58 | 0.05 | 0.065 | 33.7278 | 0.0060 | 99.3987 |
| 59 | 0.05 | 0.065 | 34.3195 | 0.0056 | 99.4368 |
| 60 | 0.05 | 0.065 | 34.9112 | 0.0053 | 99.4725 |
| 61 | 0.05 | 0.065 | 35.5030 | 0.0049 | 99.5059 |
| 62 | 0.05 | 0.065 | 36.0947 | 0.0046 | 99.5371 |
| 63 | 0.05 | 0.065 | 36.6864 | 0.0043 | 99.5663 |
| 64 | 0.05 | 0.065 | 37.2781 | 0.0041 | 99.5936 |
| 65 | 0.05 | 0.065 | 37.8698 | 0.0038 | 99.6192 |
| 66 | 0.05 | 0.065 | 38.4615 | 0.0036 | 99.6431 |
| 67 | 0.05 | 0.065 | 39.0533 | 0.0033 | 99.6655 |
| 68 | 0.05 | 0.065 | 39.6450 | 0.0031 | 99.6865 |
| 69 | 0.05 | 0.065 | 40.2367 | 0.0029 | 99.7061 |
| 70 | 0.05 | 0.065 | 40.8284 | 0.0028 | 99.7244 |

| 71 | 0.05 | 0.065 | 41.4201 | 0.0026 | 99.7416 |
|----|------|-------|---------|--------|---------|
| 72 | 0.05 | 0.065 | 42.0118 | 0.0024 | 99.7577 |
| 73 | 0.05 | 0.065 | 42.6036 | 0.0023 | 99.7728 |
| 74 | 0.05 | 0.065 | 43.1953 | 0.0021 | 99.7870 |
| 75 | 0.05 | 0.065 | 43.7870 | 0.0020 | 99.8002 |